

Version No. 5.0 Version Date: 02/08/2016

# **Bridging Study**

A Phase 2 Study Investigating Clofarabine, Cyclophosphamide and Etoposide for Children, Adolescents, and Young Adults (AYA) with Acute Leukemia and Minimal Residual Disease

**Study Chair:** Michael J. Burke, MD

Medical College of Wisconsin Department of Pediatrics

Division of Hematology/Oncology/BMT

**Study Vice Chairs:** Julie-An M. Talano, MD

Medical College of Wisconsin Department of Pediatrics

Division of Hematology/Oncology/BMT

Ehab L. Atallah, MD

Medical College of Wisconsin Department of Medicine

Division of Hematology/Oncology/BMT

**Study Committee:** Karen Sue Carlson, MD, PhD

Timothy Fenske, MD Mehdi Hamadani, MD Laura Michaelis, MD Hari Parameswaran, MD Marcelo Pasquini, MD

Gabriella Gheorghe, MD

Paul Harker-Murray, MD, PhD Michael Kelly, MD, PhD Dave Margolis, MD

Monica Thakar, MD Richard Tower, MD

**Statistician:** Raymond Hoffmann, PhD

**Additional Performance Sites:** Children's Hospital of Wisconsin

University of Wisconsin Hospital and Clinics

Nationwide Children's Hospital



# TABLE OF CONTENTS

| Section | <u>on</u> | | <b>Page</b> |
|---|---|---|---|
| Study | y Comn | nittee | 4 |
| List o | of Abbr | reviations | 6 |
| Synop | psis | | 8 |
| Protocol Revision History | | | |
| 1. | Back | ground | 13 |
| | 1.1 | High Risk ALL and AML in Children and Adults | 13 |
| | 1.2 | Overview of Cyclophosphamide and Etoposide | 14 |
| | 1.3 | Overview of Clofarabine | 14 |
| 2. | - | y Design | 19 |
| 3. | Selec | tion of Patients | 19 |
| | 3.1 | Inclusion Criteria | 19 |
| | 3.2 | Exclusion Criteria | 21 |
| 4. | _ | stration Procedures | 22 |
| | 4.1 | Registration | 22 |
| | 4.2 | Patients Who Do Not Begin Study Treatment | 22 |
| <b>5.</b> | | tment Plan | 22 |
| | 5.1 | Treatment Plan Regardless of Diagnosis | 22 |
| | 5.2 | Supportive Care Guidelines | 23 |
| | 5.3 | Duration of Therapy | 23 |
| | 5.4 | Follow-Up | 23 |
| 6. | Dose | Modification | 24 |
| | 6.1 | Clofarabine | 24 |
| | 6.2 | Cyclophosphamide | 25 |
| | 6.3 | Etoposide (VP-16) | 25 |
| <b>7.</b> | Study | y Calendar | 26 |
| | 7.1 | Standard of Care | 26 |
| 8. | Drug | Formulation and Procurement | 27 |
| | 8.1 | Clofarabine | 27 |
| | 8.2 | Cyclophosphamide | 29 |
| | 8.3 | Etoposide | 30 |
| 9. | Adve | rse Event Monitoring, Documentation, and Reporting | 31 |
| | 9.1 | Definitions | 31 |
| | 9.2 | Adverse Event Documentation | 31 |
| | 9.3 | Adverse Event Reporting Requirements | 33 |
| | 9.4 | Event Notification, Deviations, and Patient Complaints | 34 |
| 10. | Study | y Data Collection and Monitoring | 34 |
| | 10.1 | Data Management | 34 |
| | 10.2 | Case Report Forms | 35 |
| | 10.3 | Data and Safety Monitoring Plan (DSMP) | 35 |
| | 10.4 | Monitoring | 36 |
| | 10.5 | Record Retention | 36 |
| 11. | Statis | stical Considerations | 37 |
| | 11.1 | Statistic Endpoints | 37 |
| | 11.2 | Statistical Analysis | 37 |
| | 11.3 | Sample Size Justification | 37 |
| | 11.4 | Early Stopping Rule for Excessive Toxicity (pre-HCT) and | 38 |

# **Bridging Study**



# TRM (post-HCT)

| <u>Secti</u> | <u>on</u> | | <u> Page</u> |
|---|---|---|---|
| <b>12.</b> | 2. Conduct of Study | | |
| | 12.1 | Good Clinical Practice | 39 |
| | 12.2 | Ethical Considerations | 39 |
| | 12.3 | Informed Consent | 39 |
| | 12.4 | Clinical Trial Registration | 39 |
| Refe | rences | - | 40 |
| App | endix 1 - | – Eligibility Checklist | 45 |
| App | endix 2 | – Performance Status Criteria | 47 |
| App | endix 3 - | – Response Criteria | 48 |
| App | endix 4 | - Known and Expected Toxicities of Study Treatment | 49 |
| App | endix 5 | - Bridging Therapy Roadmap | 52 |



# STUDY COMMITTEE MEMBERS

| Study Chairs | |
|---|---|
| CHAIR | <b>Emergency Contact</b> |
| Michael J. Burke, MD | Children's Hospital Switchboard: |
| Associate Professor of Pediatrics | 414-266-2000 ask for Pediatric Oncologist On-Call |
| Pediatric Hematology/Oncology/BMT | |
| Medical College of Wisconsin | |
| Children's Hospital of Wisconsin | |
| 8701 Watertown Plank Road | |
| Milwaukee, WI 53226 | |
| Phone: 414-955-4198 | |
| Fax: 414-955-6543 | |
| Email: mmburke@mcw.edu | |
| VICE CHAIR | VICE CHAIR |
| Julie-An M. Talano, MD | Ehab L. Atallah, MD |
| Associate Professor of Pediatrics | Assistant Professor of Medicine |
| Pediatric Hematology/Oncology/BMT | Division of Hematology and Oncology |
| Medical College of Wisconsin | Medical College of Wisconsin |
| Children's Hospital of Wisconsin | Froedtert Memorial Lutheran Hospital |
| 8701 Watertown Plank Road | Clinical Cancer Center |
| Milwaukee, WI 53226 | 9200 W. Wisconsin Ave. |
| Phone: 414-955-4185 | Milwaukee, WI 53226 |
| Email: jtalano@mcw.edu | Phone: 414-805-4600 |
| | Email: eatallah@mcw.edu |

| Study Committee Members | |
|---|---|
| Karen Sue Carlson, MD, PhD | Timothy Fenske, MD |
| Department of Medicine – Oncology/Hematology | Department of Medicine – |
| Medical College of Wisconsin | Oncology/Hematology/BMT |
| Blood Research Institute | Medical College of Wisconsin |
| Phone: 414-805-4600 | Froedtert East Clinic |
| Email: <u>kabarker@mcw.edu</u> | Phone: 414-805-4633 |
| | Email: <u>tfenske@mcw.edu</u> |
| Gabriella Gheorghe, MD | Mehdi Hamadani, MD |
| Pediatric Medicine – Pathology | Department of Medicine – |
| Medical College of Wisconsin | Oncology/Hematology/BMT |
| Phone: 414-266-2530 | Medical College of Wisconsin |
| Email: ggheorghe@mcw.edu | Clinical Cancer Center |
| | Phone: 414-805-4600 |
| | Email: mhamadani@mcw.edu |
| Parameswaran Hari, MD | Paul Harker-Murray, MD, PhD |
| Department of Medicine – Oncology/Hematology | Pediatric Hematology/Oncology/BMT |
| Medical College of Wisconsin | Medical College of Wisconsin |
| Clinical Cancer Center | Children's Hospital of Wisconsin |
| Phone: 414-805-4602 | Phone: 414-955-4170 |
| Email: <u>phari@mcw.edu</u> | Email: <u>pharker@mcw.edu</u> |



| Study Committee Members | |
|-----------------------------------|-----------------------------------|
| Michael Kelly, MD, PhD | David Margolis, MD |
| Pediatric Hematology/Oncology/BMT | Pediatric Hematology/Oncology/BMT |
| Medical College of Wisconsin | Medical College of Wisconsin |
| Children's Hospital of Wisconsin | Children's Hospital of Wisconsin |
| Phone: 414-955-4170 | Phone: 414-955-4170 |
| Email: mekelly@mcw.edu | Email: dmargolis@mcw.edu |
| Laura Michaelis, MD | Marcelo Pasquini, MD |
| Department of Medicine – | Department of Medicine – |
| Oncology/Hematology/BMT | Oncology/Hematology/BMT |
| Medical College of Wisconsin | Medical College of Wisconsin |
| Phone: 414-805-4600 | CIBMTR |
| Email: <u>lmichaelis@mcw.edu</u> | Phone: 414-805-0700 |
| | Email: mpasquini@mcw.edu |
| Monica Thakar, MD | Richard Tower, MD |
| Pediatric Hematology/Oncology/BMT | Pediatric Hematology/Oncology/BMT |
| Medical College of Wisconsin | Medical College of Wisconsin |
| Children's Hospital of Wisconsin | Children's Hospital of Wisconsin |
| Phone: 414-955-4170 | Phone: 414-955-4170 |
| Email: mthakar@mcw.edu | Email: rtower@mcw.edu |

| Performance Site – Sub-Investigators | |
|---|---|
| Neha J. Patel, MD | Ryan Mattison, MD |
| Department of Pediatrics | University of Wisconsin Madison |
| University of Wisconsin Madison | 1111 Highland Ave. |
| 1111 Highland Ave. | 4039 Wisconsin Institute for Medical Research |
| WIMR 4 <sup>th</sup> floor North, Office # 4133 | Madison, WI 53705 |
| Madison, WI 53705 | Phone: 608-262-5697 |
| Phone: 608-263-8554 | Fax: 608-262-4598 |
| Fax: 608-265-9721 | Email: rjmattison@medicine.wisc.edu |
| Email: npatel@pediatrics.wisc.edu | |
| Susan Vear, MD | |
| Nationwide Children's Hospital | |
| 700 Children's Drive | |
| Columbus, OH 43205 | |
| Phone: 614-722-3583 | |
| Fax: 614-722-3369 | |
| Email: Susan.Vear@nationwidechildrens.org | |

| Midwest Area Research Consortium for Health (MARCH) Central Administration | |
|---|---|
| Debra Kruser | MJ Washburn |
| MARCH Director | Regional Research Networks Coordinator |
| 2112d Health Sciences Learning Center | 2112 HSLC |
| 750 Highland Ave. | 750 Highland Ave. |
| Madison, WI 53705 | Madison, WI 53705 |
| Phone: 608-262-7217 or 608-260-7633 | Phone: 608-262-7365 or 608-333-1962 |
| Email: djkruser@wisc.edu | Email: <u>mwashburn@wisc.edu</u> |



#### LIST OF ABBREVIATIONS

AE adverse event

ALL acute lymphoblastic leukemia
ALT Alanine Aminotransferase
AML acute myeloid leukemia
ANC absolute neutrophil count
APL acute promyelocytic leukemia
AST aspartate aminotransferase

AUC area under the concentration time curve

BMT bone marrow transplant

BP blood pressure BUN blood urea nitrogen

CART Therapy chimeric antigen receptor T-cell therapy CHW Children's Hospital of Wisconsin

CI confidence interval

CLL chronic lymphocytic leukemia

CNS central nervous system
CR complete remission
CrCl creatinine clearance
CRF case report forms

CRp complete remission without platelet recovery CTCAE Common Terminology Criteria for Adverse Events

CTEP Cancer Therapy Evaluation Program CTMS Clinical Trials Management System

CTO Clinical Trials Office

DEHP Bis(2-ethylhexyl) phthalate

DFS disease free survival DLT dose limiting toxicity

DSMC data safety monitoring committee
DSMP data safety monitoring plan

ECHO echocardiogram
EFS event free survival

EP European Pharmacopeia

FISH fluorescence in situ hybridisation

GFR glomerular filtration rate
GVHD graft versus host disease
GVL graft versus leukemia

HCT hematopoietic cell transplantation

HgB hemoglobin

HPLC high performance liquid chromatography
HSCT hematopoietic stem cell transplantation

HSV herpes simplex virus
IRB Institutional Review Board
LDH lactate dehydrogenase

MACC Fund Center Midwest Athletes Against Childhood Cancer Fund Center

MCW Medical College of Wisconsin MFC multiparameter flow cytometry

MRD minimal residual disease



# LIST OF ABBREVIATIONS (CONTINUED)

MTD maximum tolerated dose
MUGA multi gated acquisition scan
NOS not otherwise specified
NRM non relapse mortality

NS normal saline

ORR overall response rate
OS overall survival

PCP pneumocystis carinii pneumonia
PCR polymerase chain reaction
PI principal investigator
PR partial responsego
PVC polyvinyl chloride
RFS relapse free survival

RIC reduced intensity conditioning

SAE serious adverse event

SIRS systemic inflammatory response SRC Scientific Review Committee

UCBT umbilical cord blood transplantation

ULN upper limit of normal

UPIRSO unanticipated problems involving risks to subjects or others

USP United States Pharmacopeia

WBC white blood count



#### **SYNOPSIS**

**Study Title:** A Phase 2 Study Investigating Clofarabine, Cyclophosphamide and Etoposide for Children, Adolescents and Young Adults (AYA) with Acute Leukemia and Minimal Residual Disease

#### Phase 2

Number of Patients: 50 evaluable [25 adult (19 to 39 years) and 25 pediatric (0-18 years)]

# **Study Objectives**

# • Primary Objectives

- The effect of Clofarabine, Cyclophosphamide, and Etoposide in eliminating the presence of persistent disease without causing a significant delay of HCT due to treatment related toxicity, defined as greater than 56 days from completion of bridging therapy to start of HCT.
- The proportion of any toxicities associated with Clofarabine, Cyclophosphamide, and Etoposide

# • Secondary Objectives

- The proportion of pre-transplant chemotherapy-induced aplasia (defined as greater than 42 days after infusion of chemotherapy)
- The proportion of infectious complications following bridging therapy and before HCT
- o Treatment related mortality at Day 100 after HCT
- o One year disease-free survival after HCT
- The proportion of relapse within one year of HCT

**Treatment Plan:** Only 1 treatment course will be permitted

| Day | Agent/Procedure |
|---|---|
| Baseline | Peripheral blood draw and bone marrow aspirate (within 14 days of enrollment) |
| Day 1 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 2 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| - | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 3 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| - | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 4 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 5 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |



| Day | Agent/Proce | dure |
|---|---|---|
| Day 30* | Perform bone marrow biopsy/aspirate (*Or upon adequate blood count recover | |
| - | (ANC > 0.5 AND plt > 50,000) whichever comes first | |
| Between Day 28 & 42 | | Proceed to HCT independent of this study |

### **Study Population:**

- Diagnosis of acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) with < 5% blasts in the bone marrow (M1) by morphology and that meets one of the following criteria:
  - Flow cytometric evidence of MRD ( $\geq 0.01\%$  leukemic blasts for ALL or  $\geq 0.5\%$  leukemic blasts for AML detected in the bone marrow)

#### OR

- Molecular/cytogenetic evidence of disease (FISH or PCR methodology) performed within 14 days <u>And</u> with the intent of going on to an allogeneic hematopoietic cell transplantation (HCT) independent of this study
- Patients must have an available donor and have intention of proceeding directly to ALL-HCT after completion of 1 cycle of Bridging therapy.
- Age 0 to 39 years
- Karnofsky Performance Status  $\geq 50\%$  for patients 16 years and older and Lansky Play Score  $\geq 50$  for patients under 16 years of age (see Appendix 2)
- Patients must have a life expectancy ≥ 8 weeks as determined by the enrolling investigator
- Have acceptable organ function as defined within 7 days of study registration
  - o Renal: creatinine clearance  $\geq 60 \text{ mL/min/}1.73 \text{ m}^2$  or serum creatinine based on age/gender as follows:

| Age | Maximum Serum<br>Creatinine (mg/dl) | |
|------------------------|-------------------------------------|--------|
| | Male | Female |
| 1 month to < 6 months | 0.4 | 0.4 |
| 6 months to < 1 year | 0.5 | 0.5 |
| 1 year to < 2 years | 0.6 | 0.6 |
| 2 years to < 6 years | 0.8 | 0.8 |
| 6 years to < 10 years | 1.0 | 1.0 |
| 10 years to < 13 years | 1.2 | 1.2 |
| 13 years to < 16 years | 1.5 | 1.4 |
| ≥ 16 years | 1.7 | 1.4 |

- Hepatic: ALT < 5 x upper limit of normal (ULN) and total bilirubin  $\leq$  1.5 x upper limit of normal (ULN) for age
- o Cardiac: left ventricular ejection fraction ≥ 40% by ECHO/MUGA
- Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 7 days must have elapsed from prior chemotherapy.
- Hematopoietic Growth Factors: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.

Page 10 of 52



- Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
- Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

#### **Exclusion Criteria:**

- Acute Promyelocytic Leukemia (APL)
- Active extramedullary disease (CNS ≥ CNS2 and/or testicular leukemia) or presence of chloromatous disease
- Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anticancer therapy other than is specified in the protocol
- Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
- Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
- Known allergy to any of the agents or their ingredients used in this study
- Participating in a concomitant Phase 1 or 2 study

**Duration of Study: 2 years** 



# PROTOCOL REVISION HISTORY

| Version No. | Revision<br>Date | Summary of Changes | Consent Revised<br>Yes/No |
|---|---|---|---|
| 2.0 | 02/20/15 | Added Section 12.4 NCI trial designation number | Yes – Trial number has been added to the Consent as well |
| 3.0 | 03/20/2015 | Added Consents for Nationwide Children's and UW Madison following official deferral to MCW IRB | Yes – Added<br>consents specific to<br>Nationwide<br>Children's and UW<br>Madison |
| | | Synopsis Primary Objectives updated to provide clarification on what constitutes a delay of HCT by adding :"defined as greater than 56 days from completion of bridging therapy to start of HCT." | No |
| | | Section 2 Primary Objectives updated to provide clarification on what constitutes a delay of HCT by adding :"defined as greater than 56 days from completion of bridging therapy to start of HCT." | No |
| | | Section 3.1.1 updated to clarify and correct an inconsistency regarding inclusion criteria: flow evidence of MRD or Molecular/cytogenetic FISH or PCR evidence of disease to be performed within 14 days of enrollment | No |
| | | Section 11.1 Statistical Endpoints updated to add the definition of delay in HCT: "defined as greater than 56 days from completion of bridging therapy to start of HCT" | No |
| | | Section 11.2 Statistical Analysis correction made to SAS 9.3 changing this to SAS 9.4 | No |
| | | Section 11.3 Sample Size Justification was revised. Previous paragraph replaced with new one to strengthen the justification. | No |
| | | Section 11.4 Early Stopping Rule for Excessive Toxicity section – previous paragraph replaced with new paragraph to clarify and strengthen rationale. | No |
| 4.0 | 09/04/2015 | Page 9 Synopsis and Page 19 Section 3.1.1-<br>Eligibility Criteria changed bone marrow to be | No |



| | | performed within 14 days of enrollment (increased from within 7 days). This change did not appear in the protocol after the previous amendment and is being corrected with this amendment. This change now makes these 2 sections consistent with the table on page 26. | |
|---|---|---|---|
| | | Added Appendix 5 – Bridging therapy roadmap | No |
| | | Protocol Version number and date changed in the headers and footers to reflect the current version. | Yes – updated footers and version number – no content changes |
| | | Table of contents updated. | No |
| 5.0 | 02/08/2016 | Headers and Footers updated with new version number and date Page 5 Performance Site Sub Investigators: Replaced Robyn Dennis, MD with Susan Vear, MD at Nationwide Children's Hospital | Yes- updated footers with new protocol version number and date. All Assents section E2 replaced Robyn Dennis, MD with Susan Vear, MD as contact for Nationwide Children's Hospital All Consents Section D5 replaced Robyn Dennis, MD with Susan Vear, MD as contact for Nationwide Children's Hospital Consents Section D5 replaced Robyn Dennis, MD with Susan Vear, MD as contact for Nationwide Children's Hospital |



#### 1. BACKGROUND

# 1.1 High Risk ALL and AML in Children and Adults

Acute lymphoblastic leukemia (ALL) and acute myeloid leukemia (AML) remain two of the most common forms of leukemia diagnosed in both children and adults, as well as two of the most common hematological diseases for which allogeneic hematopoietic cell transplantation (HCT) is currently used.<sup>12</sup> There is mounting evidence to support that for patients in hematological remission, the presence of minute amounts of leukemia (known as minimal residual disease (MRD)), identified immediately prior to HCT is associated with higher rates of ALL and AML relapse following HCT.<sup>1-11</sup> Therefore we hypothesize that transplant outcomes can be improved by reducing pre-HCT disease burden by attaining a pre-HCT MRD negative state. We designed this protocol to test the combination of clofarabine, cyclophosphamide and etoposide, which are known active agents in the treatment of lymphoid and myeloid hematologic malignancies, in their ability to both lower MRD and improve post-HCT outcomes for patients with ALL/AML who are in morphological remission but have evidence of MRD pre-HCT.

Impact of MRD Positive Disease Prior to HCT: Patients with acute leukemia and submorphologic disease at the time of conditioning are at high risk of relapse following HCT. Recent studies have demonstrated that even low levels of MRD (> 0.01% abnormal blasts by multi-parameter flow cytometry, MFC) after aggressive re-induction therapy portends a relatively poor outcome in relapsed ALL patients, including those who proceed to HCT. Foster et al. recently reported 116 pediatric patients who were in morphologic remission and underwent MRD evaluation with multi-parameter flow cytometry (MFC) prior to ablative transplant for ALL. For the group as a whole, the EFS for MRD positive and negative patients was 11% and 58% respectively, (p < 0.001).<sup>3</sup>

Likewise, the BFM Study Group has also evaluated the impact of MRD prior to HCT for relapsed ALL using a PCR-based assay. Their multivariate Cox regression analysis revealed MRD as the only independent parameter predictive for EFS (p < 0.006).

MRD identified prior to HCT for AML portends a poor prognosis in both pediatric and adult patients. <sup>13-16</sup> In a report by Walter et al. 99 pediatric and adult patients with AML receiving a HCT in CR1 were evaluated for pre-HCT MRD using MFC with any detectable MRD defined as MRD-positive. <sup>13</sup> The 2-year EFS for MRD-positive patients was 9% with a relapse rate of 64.9% compared to 74.8% and 17.6% in MRD-negative patients respectively. The multivariate analysis identified pre-HCT MRD as a significant risk factor for both overall mortality (HR 4.05 95% CI 1.90-8.62, p < 0.001) and relapse (HR 8.49 95% CI 3.67-19.65, p < 0.001). In another analysis reporting a larger group of pediatric and adult patients with AML (n=253) receiving HCT in CR1 or CR2, OS (HR 2.61, 95% CI 1.62-4.20, p < 0.001), DFS (HR 3.74, 95% CI 2.38-5.87, p < 0.001), and relapse (HR 4.90, 95% CI 2.87-8.37, p < 0.001) were all significantly worse for patients identified as MRD-positive MFC (≥ 0.1% blasts), compared to MRD-negative patients in multivariate cox regression model. <sup>14</sup>



Numerous monitoring techniques such as MFC, monitoring of known cytogenetic abnormalities, and molecular abnormalities such as NPM-1 and WT-1 have identified MRD in this patient population. <sup>14,17,18</sup> One of the larger recent studies investigating the impact of MRD on post-transplant outcomes for AML patients evaluated 88 patients with morphologic CR, 24 of which had MRD by MFC, who went on to receive a myeloablative transplant. Survival and relapse were strongly associated with absence or presence of MRD. Specifically, two year overall survival was 30.2% (range 13-49%) for the MRD-positive patients compared with 76.6% (64.4-85.1%) for those who were MRD-negative. Two year estimates of relapse also correlated with MRD status with rates of 65% in those who were MRD-positive compared with 17.6% in those MRD-negative. These data highlight the significance of MRD on post-transplant relapse and the need for improved therapy.

Investigators at the University of Minnesota analyzed 97 adult AML patients; 14 had detectable MRD prior to allogeneic donor HCT. Overall survival and disease free survival were markedly worse in MRD-positive patients receiving RIC compared to MRD-negative cohort. This research also investigated impact of pre-transplant MRD (assessed by MFC) in adults and children with ALL prior to umbilical cord blood transplantation. Patients with MRD-positive prior to UCBT had a greater incidence of relapse at 2-years (30% (95% CI: 4-56%) and lower 3-year disease-free survival (DFS) (30%; 95% CI 7-58%) compared to MRD-patients (relapse 16% (95% CI: 8-25%: p=0.05 and DFS 55%; 95% CI: 43-66%; p=0.02). These data suggest that in the majority of patients with residual leukemia at the time of HCT, neither the preparative regimen, nor the GVL effect of the allograft is sufficient to prevent relapse. Thus, methods to eliminate persistent leukemia that have low toxicity profiles and can serve as a "bridge" to transplant are needed.

## 1.2 Overview of Cyclophosphamide and Etoposide

The combination of the alkylating agent cyclophosphamide with the topoisomerase II inhibitor etoposide has been a common re-induction therapy for relapse/refractory acute leukemia. These two agents have been used in combination in a number of recent studies through the Children's Oncology Group (COG) in both AALL01P2 for relapse B-Precursor ALL as well as the Infant ALL study CCG 1953 with limited toxicities. In addition the combination has been evaluated in adult patients with relapsed/refractory AML. Of the 34 patients enrolled, 27 received etoposide 3 gm/m² by continuous infusion over 48-72 hours, immediately followed by cyclophosphamide 50 mg/kg iv over 3 hours daily for 3 or 4 days (150-200 mg/kg total dose). The other seven patients received a lower etoposide dose, 1.8–2.4 gm/m² over 48-72 hours followed by cyclophosphamide 50 mg/kg IV over 3 hours for 3 or 4 days. The complete remission rate and treatment related mortality was 32% and 18% respectively. These results compare favorably to other salvage regimens used in the treatment of patients with relapsed refractory AML. Recently they have been shown to be synergistic with the relatively new purine nucleoside analogue clofarabine.

#### 1.3 Overview of Clofarabine

Clofarabine (2-chloro-9-[2'-deoxy-2'-fluoro-β-D-arabinofuranosyl]adenine; Cl-F-ara-A;



CAFdA) is a rationally designed, second generation purine nucleoside analogue. Clofarabine was designed as a hybrid molecule to overcome the limitations and incorporate the best qualities of both fludarabine (F-ara-A) and cladribine (2-CdA, CdA) both of which are currently approved by various regulatory authorities for treatment of hematologic malignancies. Because clofarabine has a chloro-group at the 2-position of adenine, its chemical structure is more closely related to 2-CdA than to F-ara-A.<sup>26</sup> Halogenation at the 2-position of adenine renders this class of compounds resistant to intracellular degradation by the enzyme adenosine deaminase. Substitution of a fluorine at the C-2'-position of the arabinofuranosyl moiety of clofarabine increases its stability in gastric acid<sup>27</sup> and decreases its susceptibility to phosphorolytic cleavage by the bacterial enzyme Escherichia coli purine nucleoside phosphorylase in the gastrointestinal tract, 28 both of which may lead to enhanced oral bioavailability. Clofarabine was approved in December 2004 by the United States Food and Drug Administration (US FDA) for the treatment of pediatric patients with relapsed or refractory acute lymphoblastic leukemia (ALL) after at least 2 prior regimens based on the induction of complete responses.

**Mechanism of Action:** The precise mechanism of action of clofarabine on dividing and non-dividing cells is unknown. Like the other nucleoside analogues (cytarabine, ara-A [vidarabine], cladribine, fludarabine), clofarabine must be converted to the 5'triphosphate form by deoxycytidine kinase (dCK) to be active within cells. Clofarabine is more efficient as a substrate for purified recombinant dCK, exceeding cladribine and the natural substrate, deoxycytidine.<sup>29</sup> Evidence suggests that the primary cytotoxic effect of clofarabine is due to its inhibition of DNA synthesis. The triphosphate form of clofarabine is an inhibitor of both DNA polymerase α and ribonucleotide reductase.<sup>30</sup> These effects lead to depletion of intracellular deoxynucleotide triphosphate pools, and inhibition of elongation of DNA strands during synthesis. 26 With respect to inhibition of ribonucleotide reductase, clofarabine and cladribine are superior to fludarabine.<sup>30</sup> With respect to inhibition of DNA polymerase α, clofarabine and fludarabine are similar and both are superior to cladribine.<sup>28</sup> Thus, in comparison to cladribine and fludarabine. clofarabine more completely inhibits both ribonucleotide reductase and DNA polymerase  $\alpha$ , versus one or the other. Clofarabine is active in non-dividing cells and in cells with a low proliferation rate. Clofarabine has been shown to disrupt the integrity of mitochondria in primary chronic lymphocytic leukemia (CLL) cells. The damage leads to release of pro-apoptotic mitochondrial factors.<sup>31</sup> These effects are postulated to induce apoptosis in indolent, non-dividing CLL cells. This result was not seen with fludarabine and may explain, at least in part, the enhanced cytotoxicity of clofarabine<sup>30</sup> though the physiologic and clinical implications of these observations remain uncertain and under continued investigation.

## **Experience With Clofarabine in Pediatric Leukemia**

**Phase 1 Clofarabine Studies:** In the initial Phase 1 study in pediatric patients with hematologic malignancies, 25 patients were treated in cohorts of escalating doses up to 70 mg/m<sup>2</sup>, a dose at which 1 patient had grade 4 hyperbilirubinemia and grade 3 elevated transaminases, and 1 had a grade 3 skin rash. The MTD was determined to be 52 mg/m<sup>2</sup>.<sup>27</sup> Of the 13 patients treated at 52 mg/m<sup>2</sup>, grade 2 to grade 3 increases in bilirubin and liver transaminases were observed. A total of 5 patients achieved a CR and 3 achieved a PR for an overall response rate of 32%. Clofarabine plasma concentrations



were generally lower in the pediatric population than the adult population when administered the same dose, but there did not appear to be much difference in intracellular clofarabine triphosphate concentrations. Thus, the MTD and the recommended Phase 2 dose was determined to be 52 mg/m² and the recommended Phase 2 dose. The Phase 1 studies in pediatric patients with hematologic malignancies led to the initiation of 2 parallel Phase 2 trials in 2002 for patients with either relapsed or refractory ALL or relapsed or refractory AML.<sup>29</sup>

Both studies evaluated clofarabine 52 mg/m<sup>2</sup>. In the 61 patients enrolled in the relapsed or refractory ALL study (61% males: 39% females, 1 to 20 years old), the overall remission rate (CR + CRp) was 20%; 30% (18/61) of patients showed a response (7CR, 5CRp, 6PR). Responses were noted in 15 of 50 (30%) patients with Blineage ALL, 2 of 6 (33%) with T-cell ALL. Responders received a median of 3 prior induction regimens; 50% (9/18) had prior HSCT and 50% (9/18) were refractory to the preceding induction regimen. Response rate in refractory patients was 26% (9/35). After clofarabine treatment, 10 patients proceeded to transplant (including 8 responders). Six of 10 patients who received a transplant were alive at last follow up (survival range: 30.1+ to 145.1+ weeks). Response duration in 6 patients with CR or CRp who did not receive a transplant ranged from 4.3 to 58.6 weeks; 2 patients maintained CR for 47.9 and 58.6 weeks after clofarabine therapy. Median overall survival for the patients who achieved at least a PR was 66.6 weeks compared to 12.9 weeks for all patients.<sup>29</sup> In 42 pediatric patients with relapsed or refractory AML, the response rate was 26% (1 CRp, 10 PR). Responders had received a median of 2 prior induction regimens, 36% (4/11) had prior HCT and 55% (6/11) patients were refractory to the preceding induction regimen. Response rate in refractory patients was 21% (6/28). One patient who had received 5 prior induction regimens achieved CRp. 13 (31%) patients (1CRp, 6PR, 3NE, 3TF) underwent HSCT after completing clofarabine therapy, 5 of whom were alive at last follow-up (survival range: 62.7+ to 160.1+ weeks). Many patients proceeded to HSCT as soon as a donor was identified without waiting for the patient to go into remission, making remission difficult to assess. Median overall survival for patients who achieved at least a PR was 32.1 weeks compared to 23.4 weeks for all patients.<sup>32</sup>

Among the 113 pediatric patients with ALL and AML, the most frequently reported drug-related AEs were vomiting (66% ALL and 65% AML) and nausea (58% ALL and 70% AML). Other drug-related AEs reported by at least 10% of the pediatric patients overall included febrile neutropenia (31% ALL and 28% AML), pyrexia (21% ALL and 26% AML), pruritus NOS (24% ALL and 20% AML), dermatitis NOS (24% ALL and 17% AML), headache NOS (18% ALL and 35% AML), diarrhea NOS (21% ALL and 22% AML), anxiety (16% ALL and 7% AML), fatigue (15% ALL and 13% AML), mucosal inflammation NOS (16% ALL and 15% AML), and flushing (12% ALL and 11% AML). Anorexia occurred in 12% ALL and 9% AML and palmar-plantar erythrodysesthesia syndrome in 12% ALL and 9% AML.

**Phase 2 Clofarabine Studies:** A Phase 2 trial of clofarabine in combination with cyclophosphamide and etoposide in pediatric patients with refractory/relapsed acute lymphoblastic leukemia was recently reported by Hijiya et al.<sup>25</sup> The efficacy and safety of intravenous clofarabine 40 mg/m<sup>2</sup> per day, cyclophosphamide 440 mg/m<sup>2</sup> per day, and etoposide 100 mg/m<sup>2</sup> per day for 5 consecutive days in pediatric patients with



refractory or relapsed ALL was evaluated in this Phase 2 study. The primary endpoint was overall response rate (complete remission [CR] plus CR without platelet recovery [CRp]). Among the 25 patients (median age, 14 years; pre-B cell ALL, 84%; ≥ 2 prior regimens: 84%; refractory to previous regimen: 60%), the overall response rate was 44% (7 CR, 4 CRp) with a 67.3-week median duration or remission censored at last follow-up. Most patients proceeded to alternative therapy, and 10 patients (40%) received HCT. Six patients (24%) died because of treatment-related adverse events associated with infection, hepatotoxicity, and/or multi-organ failure. The study protocol was amended to exclude patients with prior hematopoietic stem cell transplantation after 4 of the first 8 patients developed severe hepatotoxicity suggestive of veno-occlusive disease. No additional cases of veno-occlusive disease occurred.

# **Experience With Clofarabine in Adult Patients**

Clofarabine activity has been evaluated in children and adults with acute leukemia and found to have no difference in activity between these two age groups.<sup>33</sup> Based on this finding as well as the known clinical activity using clofarabine in relapsed pediatric ALL and AML,<sup>25,29</sup> it is reasonable to further evaluate the clinical efficacy of clofarabine in combination with chemotherapy in adult patients with acute leukemia.

Phase 1 Clofarabine Studies: Clofarabine was evaluated in a Phase 1 study in patients with both hematologic malignancies and solid tumors. In patients with solid tumors, the starting dose level was 15 mg/m<sup>2</sup> daily for 5 days. Grade 4 myelosuppression occurred and the clofarabine dose was reduced by several dose levels with the MTD defined at 2 mg/m<sup>2</sup> in patients with solid tumors. In patients with leukemia, the starting dose level was 7.5 mg/m<sup>2</sup>. This dose was escalated by several dose levels until 55 mg/m<sup>2</sup> was achieved. At the 55 mg/m<sup>2</sup> dose level, grade 3 hepatic toxicity was observed in 2 of 4 patients, which caused dose de-escalation to 40 mg/m<sup>2</sup> and became the recommended Phase 2 dose. This cohort was expanded to include 12 patients. Of the 12 patients treated at 40 mg/m<sup>2</sup>, 2 patients achieved CR (1 AML and 1 ALL) suggesting some efficacy and safety at this dose level in patients with acute leukemia Based on in vitro data suggesting synergism between clofarabine and cyclophosphamide, Karp et al designed a Phase 1study with escalating doses of both agents<sup>34</sup>. Of the 18 patients enrolled, 12 and 6 had relapsed or refractory AML and ALL respectively. The median age was 51. Dose Level 1 was cyclophosphamide 200 mg/m<sup>2</sup> on Days 0 and 1, cyclophosphamide 400 mg/m<sup>2</sup> on Days 2, 3, and 8-10, and clofarabine 20 mg/m<sup>2</sup> Days 1-3 and 8-10. The total cyclophosphamide and clofarabine dose was 2400 mg/m<sup>2</sup> and 120 mg/m<sup>2</sup> respectively. In our study, the total cyclophosphamide and clofarabine dose is 1500 mg/m<sup>2</sup> and 100 mg/m<sup>2</sup> respectively. At that dose level, 2 of the 6 patients experienced prolonged bone marrow suppression which led to the reduction of the clofarabine dose to 10 mg/m<sup>2</sup>. At this dose level, one death occurred at Day 14 and that cohort was expanded to include 12 patients and was defined as the DLT. Overall 4 patients died on the study, 2 in each dose cohort. The median time to bone marrow recovery was decreased from 45 days to 35 days from Dose Level 1 to Dose Level 0. Of the 12 patients enrolled at Dose Level 0, 3 patients achieved a CR suggesting activity of this combination in adult relapsed/refractory leukemia.

**Phase 2 Clofarabine Studies:** A Phase 2 study enrolled 116 newly diagnosed AML



patients with a median age of 71 years.<sup>35</sup> Unfavorable cytogenetics were present in 55%. Clofarabine at 30 mg/m<sup>2</sup> IV was administered daily for 5 days for induction followed by 20 mg/m<sup>2</sup> for 5 days as consolidation. The ORR was 46% with 38% of patients achieving a CR or CRp. The median overall survival for all patients, patients in CR/CRp and those in CR was 41, 59 and 72 weeks respectively. Overall clofarabine was well tolerated with a 60-day mortality rate of 16% (from any cause).

## **Study and Dose Rationale**

The safety profile of clofarabine appears acceptable within the target populations studied to date in the clinical studies summarized above. Clofarabine has demonstrated anticancer activity through inhibition of DNA synthesis and repair, induction of apoptosis, and possibly through other mechanisms. Numerous responses have been observed after treatment with clofarabine in heavily pre-treated relapsed/refractory patients with ALL or AML. Additionally there have been responses in several adult studies of lower dose clofarabine in combination with a variety of agents. The patient population selected, MRD positive prior to transplantation would be an ideal patient population to investigate the role of a "bridge" chemotherapy combination prior to HCT and potentially improve the event-free survival (EFS) of this group of patients who historically have had inferior outcomes but are ineligible for most current relapsed studies.

# Experience With Clofarabine/Cyclophosphamide/Etoposide as Bridging Therapy in Pediatric ALL

Investigators at the University of Minnesota have been using this combination of lower dose clofarabine and cyclophosphamide with etoposide as "bridging therapy" for patients with B-precursor ALL who were in a morphologic remission (< 5% leukemia blasts in the marrow) but with evidence of MRD (> 0.01% leukemia blasts) via flow cytometry and awaiting HCT. To date, they have treated three pediatric patients with this regimen and in all three achieved MRD reduction (2/3 becoming MRD-negative) after a single course of therapy and experienced no Grade III/IV toxicities with both rapid neutrophil and platelet recovery. All three patients successfully proceeded to HCT after completion of this bridging therapy without further delay or toxicity and have experienced no increase in post-HCT toxicity.

Based on the success using this clofarabine-based regimen at the University of Minnesota, five additional patients were treated at four pediatric centers across the US, all with MRD-positive ALL (ages ranging 23 months to 20 years). All 5 patients had reduction in MRD after a single course of therapy with 4/5 achieving MRD-negativity. All 5 patients proceeded to HCT with 4/5 alive and free of disease at the time of this report and one case of TRM.

Reporting the results of all 8 patients treated with this bridging regimen across all centers provides 1-year EFS of 44% (95% CI 6-81) with two relapses occurring. One relapse occurred in a patient with Philadelphia chromosome positive B-ALL who received the bridging therapy, but remained with persistent MRD prior to HCT, which incidentally was a reduced intensity conditioning regimen and the patient's 2<sup>nd</sup> HCT. The second relapse occurred in a patient with *MLL* gene rearrangement who achieved



MRD-negativity post-bridging therapy but subsequently relapsed 106 days post-HCT. This patient then received another course of the clofarabine-based bridging regimen resulting in elimination of his disease becoming MRD-negative  $(4\% \rightarrow < 0.01\%$  by flow cytometry) and proceeded to chimeric antigen receptor T-cell (CART) therapy.

## **Experience With Clofarabine as Bridging Therapy in Adult Patients With AML**

Clofarabine when given immediately prior to HCT was found to be safe in the setting of haploidentical HCT. In a study by Tischer et al, 18 patients with relapsed leukemia were enrolled, 15 having the diagnosis of AML.<sup>39</sup> All patients had active leukemia at time of HCT and received cytoreductive chemotherapy with clofarabine at a dose of 30 mg/m<sup>2</sup> IV over 5 days followed by 3 days of rest prior to starting their HCT conditioning regimen. Conditioning consisted of five doses of fludarabine at 30 mg/m<sup>2</sup>/day IV and two doses of cyclophosphamide at 14.5 mg/kg/day IV. The estimated OS, RFS and NRM was 55.5%, 39% and 23% respectively. Five patients died from NRM with 4 patients dying from infectious complications and one patient dying from liver toxicity, and GVHD.

#### 2. STUDY DESIGN

This is a Phase 2 study designed for the purpose of estimating various parameters surrounding the efficacy of Clofarabine, Cyclophosphamide and Etoposide in eliminating minimal residual disease (MRD) in acute leukemia patients otherwise in remission and without causing significant delay of HCT due to treatment related toxicity. A single course of "bridge" chemotherapy is given prior to the transplant procedure as an approach to improved disease-free survival in a patient group who historically has had inferior outcomes.

The following parameters will be monitored.

#### **Primary Objectives**

- The effect of Clofarabine, Cyclophosphamide and Etoposide in eliminating the presence of MRD without causing a significant delay of HCT due to treatment related toxicity, defined as greater than 56 days from completion of bridging therapy to start of HCT
- The proportion of any toxicities associated with Clofarabine, Cyclophosphamide and Etoposide

## **Secondary Objectives**

- The proportion of pre-transplant chemotherapy-induced aplasia (defined as greater than 42 days after infusion of chemotherapy)
- The proportion of infectious complications following bridging therapy and before HCT
- Treatment–related mortality at Day 100 after HCT
- One year disease-free survival after HCT
- The proportion of relapse within one year of HCT



#### 3. SELECTION OF PATIENTS

Study entry is open to patients regardless of gender or ethnic background. While there will be every effort to seek out and include females and minority patients, the patient population is expected to be no different than that of other acute leukemia studies at the Medical College of Wisconsin.

#### 3.1 Inclusion Criteria

- **3.1.1** Diagnosis of ALL or AML with < 5% blasts in the bone marrow (M1) by morphology and that meets one of the following criteria:
  - a. Flow cytometric evidence of MRD ( $\geq 0.01\%$  leukemic blasts for ALL or  $\geq 0.5\%$  leukemic blasts for AML detected in the bone marrow)

#### OR

- b. Molecular/cytogenetic evidence of disease (FISH or PCR methodology) performed within 14 days
- **AND** with the intent of going on to an allogeneic hematopoietic cell transplantation (HCT) independent of this study
- **3.1.2** Patients must have an available donor and have intention of proceeding directly to ALL-HCT after completion of 1 cycle of Bridging therapy.
- **3.1.3** Age 0 to 39 years
- **3.1.4** Karnofsky Performance Status  $\geq 50\%$  for patients 16 years and older and Lansky Play Score  $\geq 50$  for patients under 16 years of age (see Appendix 2)
- 3.1.5 Patients must have a life expectancy  $\geq 8$  weeks as determined by the enrolling investigator
- **3.1.6** Have acceptable organ function as defined within 7 days of study registration:

**Renal:** creatinine clearance  $\geq 60 \text{ mL/min/}1.73\text{m}^2 \text{ or}$  serum creatinine based on age/gender as follows:

| | Maximum Serum | |
|------------------------|--------------------|--------|
| Age | Creatinine (mg/dl) | |
| | Male | Female |
| 1 month to < 6 months | 0.4 | 0.4 |
| 6 months to < 1 year | 0.5 | 0.5 |
| 1 year to < 2 years | 0.6 | 0.6 |
| 2 years to < 6 years | 0.8 | 0.8 |
| 6 years to < 10 years | 1.0 | 1.0 |
| 10 years to < 13 years | 1.2 | 1.2 |



| Age | Maximum Serum<br>Creatinine (mg/dl) | |
|------------------------|-------------------------------------|-----|
| 13 years to < 16 years | 1.5 | 1.4 |
| ≥ 16 years | 1.7 | 1.4 |

<u>Hepatic</u>: ALT < 5 x upper limit of normal (ULN) and total bilirubin  $\le 1.5$  x upper limit of normal (ULN) for age

<u>Cardiac:</u> left ventricular ejection fraction ≥ 40% by ECHO/MUGA

**3.1.7** Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 7 days must have elapsed from prior chemotherapy.

<u>Hematopoietic Growth Factors</u>: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.

- **3.1.8** Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
- **3.1.9** Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

#### 3.2 Exclusion Criteria

- **3.2.1** Acute Promyelocytic Leukemia (APL)
- **3.2.2** Active extramedullary disease (CNS  $\geq$  CNS2 and/or testicular leukemia) or presence of chloromatous disease
- **3.2.3** Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy other than is specified in the protocol
- **3.2.4** Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
- 3.2.5 Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.



- **3.2.6** Known allergy to any of the agents or their ingredients used in this study
- **3.2.7** Participating in a concomitant Phase 1 or 2 study

#### 4. REGISTRATION PROCEDURES

Registration will occur after eligibility is confirmed and the patient/parent has signed the subject consent, but before any treatment has been administered.

The eligibility checklist will be completed at the time of study enrollment.

# 4.1 Registration

Upon completion of the screening evaluation, eligibility confirmation and obtaining written consent, the patient will be registered in the study file by the Department of Pediatrics Division of Hematology/Oncology/BMT MACC Fund Center Clinical Trials Office (CTO). When the Research Electronic Data Capture (REDCap) Database is fully functioning for this study, the MARCH Consortium will use this program for patient registration.

# 4.2 Patients Who Do Not Begin Study Treatment

If a patient is registered on the study, and is later found not able to begin the planned study treatment, for whatever reason, the patient will be removed from study and treated at the physician's discretion. Study data will be collected until the time of study removal. The reason for removal from study will be clearly indicated on the case report forms.

If a patient begins treatment, and then is discontinued for whatever reason, the patient must be followed per Section 5.4.

# 5. TREATMENT PLAN

The administration of the study drugs will follow institutional drug and supportive care guidelines. Refer to Section 5.2 for additional therapy based on specific disease features.

Only 1 treatment course is permitted.

## 5.1 Treatment Plan Regardless of Diagnosis

| Day | Agent/Procedure |
|---|---|
| Baseline | Peripheral blood draw and bone marrow aspirate (within 14 days of enrollment) |
| Day 1 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 2 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosphamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |



| Day | Agent/Proce | dure |
|---|---|---|
| Day 3 | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by | |
| | | 0 mg/m <sup>2</sup> IV over 2 hours followed by |
| | | amide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 4 | | Clofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Etoposide 10 | 0 mg/m <sup>2</sup> IV over 2 hours followed by |
| | | amide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 5 | | ofarabine 20 mg/m <sup>2</sup> IV over 2 hours followed by |
| - | | le 100 mg/m <sup>2</sup> IV over 2 hours followed by |
| | Cyclophosph | bhamide 300 mg/m <sup>2</sup> IV as a 30-60 minute infusion |
| Day 30* | Perform bone marrow biopsy/aspirate (*Or upon adequate blood count recover | |
| | (ANC > 0.5 AND plt > 50,000) whichever comes first | |
| Between Da | n Day 28 & 42 Proceed to HCT independent of this study | |

Pretreatment stress doses of steroids (i.e. hydrocortisone 50-100 mg/m²/dose IV daily) during clofarabine administration for prophylaxis against SIRS is allowed on study.

A bone marrow evaluation to determine study response and remission status will be performed on study Day 30 or upon adequate blood count recovery (ANC > 0.50 and platelet > 50,000), whichever occurs first. If the marrow is hypocellular and without evidence of normal tri-lineage hematopoiesis the marrow should be repeated at Day 42.

# **5.2** Supportive Care Guidelines

All supportive measures consistent with optimal patient care will be given throughout the study.

**Venous Access:** A central venous access device, preferably a double lumen, is strongly recommended for this study.

Anti-emetics will be used according to standard medical practice. Growth factor use is allowed on this study.

**Antimicrobial Prophylaxis:** Patients should be placed on standard of care prophylaxis during this time period at the discretion of the treating physician according to institutional guidelines for PCP, HSV, bacterial and fungus.

#### 5.3 **Duration of Therapy**

Treatment will be limited to one course. Patients will receive protocol therapy unless:

- Patient withdraws consent or is non-compliant
- Disease progression
- Inter-current illness that prevents further administration of treatment
- Unacceptable toxicity

# 5.4 Follow-Up

All patients, including those who discontinue protocol therapy early, will be followed



for 60 days from the first dose of study drug or until the start of the transplant prep regimen (or other therapy), whichever occurs earlier.

For patients who go on to transplant (the intent of this study), routine outcomes (treatment related mortality, disease free survival) will be abstracted from the Blood and Marrow Transplantation (BMT) database through the 3<sup>rd</sup> year post-transplant follow-up.

#### 6. DOSE MODIFICATION

The intent of this study design is for all patients to receive and complete one course of therapy. Patients who exhibit signs of disease progression or experience an unacceptable toxicity will be discontinued from treatment.

There will be no dose delays or dose reductions of study drugs for hematologic toxicity during Consolidation "Bridging" therapy (Day 1 through Day 30); however, prolonged hematopoietic recovery or bone marrow aplasia during the first 42 days may meet a study stopping rule per Section 11.4.

#### 6.1 Clofarabine

**Cardiac Dysfunction (Grade 3-4):** Discontinue clofarabine administration for Grade 3-4 left ventricular systolic dysfunction.

**Hyperbilirubinemia (Grade 3-4):** Hold clofarabine administration if Grade 3 or higher increase in bilirubin is noted. If the patient's condition stabilizes and organ function has returned to baseline, clofarabine administration may be continued at a 25% dose reduction.

**Pancreatitis** (Grade 3-4): Discontinue clofarabine in the presence of hemorrhagic pancreatitis or severe pancreatitis. In the case of mild pancreatitis, clofarabine should be held until symptoms and signs subside, and amylase levels return to normal and then resumed at a 25% dose reduction.

**Renal Dysfunction (Grade 3-4):** Hold clofarabine administration if Grade 3 or higher increase in creatinine is noted. Adjust clofarabine as follows:

- GFR/CrCl 30 < 60 mL/min/1.73 m<sup>2</sup>: Decrease dose by 50%
- GFR/CrCl < 30 mL/min/1.73 m<sup>2</sup>: Do **NOT** administer clofarabine. Resume only when ≥ 30 mL/min/1.73 m<sup>2</sup>

Systemic Inflammatory Response (SIRS)/Capillary Leak Syndrome: Hold clofarabine administration if signs of SIRS develops (tachypnea or other evidence of respiratory distress, unexplained hypotension and/or unexplained tachycardia). Although clofarabine has been associated with systemic inflammatory response, other causes of SIRS, such as infection, should be investigated. If the patient's condition stabilizes or improves, clofarabine administration may be continued at a 25% dose reduction with the addition of pretreatment stress doses of steroids (e.g. hydrocortisone 50-100 mg/m²/dose IV daily during clofarabine administration).



# 6.2 Cyclophosphamide

**Hematuria:** Omit in the presence of macroscopic hematuria. If there is a history of previous significant hematuria, hydrate before cyclophosphamide until specific gravity is < 1.010 and hydrate at 125 mL/m²/hr for 24 hours after dose. Monitor for adequate urine output as per institution guidelines. Give IV mesna at a total dose that is 60% of the cyclophosphamide dose divided to 3 doses (i.e. if the cyclophosphamide dose is 1000 mg/m², the total mesna dose is 600 mg/m² or 200 mg/m²/dose). Give the first mesna dose 15 minutes before or at the same time as the cyclophosphamide dose and repeat 4 and 8 hours after the start of cyclophosphamide. This total daily dose of mesna can also be administered as IV continuous infusion. The continuous infusion should be started 15-30 minutes before or at the same time as cyclophosphamide and finished no sooner than 8 hours after the end of cyclophosphamide infusion.

**Renal Dysfunction:** If creatinine clearance or radioisotope GFR is < 10 mL/min/1.73 m<sup>2</sup>, reduce dose of cyclophosphamide by 50%. Prior to dose adjustment of cyclophosphamide, the creatinine clearance should be repeated with good hydration.

# 6.3 Etoposide (VP-16)

**Allergic Reaction:** Pre-medicate with diphenhydramine (1-2 mg/kg slow IV push, maximum dose is 50 mg). If symptoms persist, add hydrocortisone 100-300 mg/m<sup>2</sup>. Continue to use premedication before etoposide in future. Also consider substituting an equimolar amount of etoposide phosphate, in the face of significant allergy and/or hypotension. Etoposide phosphate is a water soluble prodrug that does not contain polysorbate 80 and polyethyleneglycol, the solubilizing agent in etoposide that may induce allergic reactions and hypotension. Etoposide phosphate is rapidly converted to etoposide *in vivo* and provides total drug exposure, as represented by AUC (0-infinity) that is statistically indistinguishable from that measured for etoposide at equimolar doses.

**Hypotension:** If diastolic or systolic blood pressure (BP) falls 20 mmHg during infusion, reduce infusion rate by 50%. Start a simultaneous infusion of NS 10 mL/kg if BP fails to recover or falls further. Stop infusion if BP does not recover, continue NS. If the patient has had any episode of hypotension, prehydrate with 0.9% NaCl at 10 mL/kg/hr for 2 hours prior to any subsequent infusion.

**Renal Insufficiency:** If renal function decreases, adjust etoposide as follows: CrCl 10-50 mL/min/1.73 m<sup>2</sup>, decrease dose by 25%; if CrCl < 10 mL/min/1.73 m<sup>2</sup>, decrease dose by 50%.

**Hyperbilirubinemia:** If direct bilirubin is > 2 mg/dL, decrease dose by 50%. If direct bilirubin is > 5 mg/dL, hold etoposide.



# 7. Study Calendar

## 7.1 Standard of Care

| Evaluations | Pre- | Day | Day | Day |
|---|---|---|---|---|
| | Study | 1-5 | 6-29 | 30-60 <sup>4</sup> |
| Clinical history | X | | | |
| Physical exam | X | X | Weekly | Weekly |
| Vital exam | X | X | Weekly | Weekly |
| Weight | X | | Weekly | Weekly |
| Height | X | | | |
| Performance status | X | | Weekly | Weekly |
| Adverse event, toxicity notation | X | X | Weekly | Weekly |
| La | boratory | | | |
| WBC, Hgb, platelets, diff | X | X | Twice Weekly | Twice Weekly |
| Electrolytes including Ca++, PO4, Glucose | X | X | Weekly | Weekly |
| BUN, Creatinine, ALT, AST, LDH, | X | X | Weekly | Weekly |
| Alkaline Phosphatase, bilirubin | | | | |
| Albumin and Total Protein | X | | | |
| Serum amylase and lipase | X | | | |
| Urinalysis | X | | | |
| Creatinine clearance <sup>1</sup> | X | | | |
| Echocardiogram/MUGA | X | | | |
| Pregnancy test <sup>2</sup> | X | | | |
| Bone marrow aspirate (within 14 days of | X | | | $X^3$ |
| enrollment for pre-study sample) <sup>6</sup> | | | | |
| Lumbar puncture <sup>5</sup> | X | | | |
| Treatment | | | | |
| Clofarabine | | Daily | | |
| Etoposide | | Daily | | |
| Cyclophosphamide | | Daily | | |

Optional for eligibility, see Section 3.5

<sup>&</sup>lt;sup>2</sup> For females of childbearing potential only

<sup>&</sup>lt;sup>3</sup> A bone marrow evaluation to determine study response and remission status will be performed on study Day 30 or upon adequate blood count recovery (ANC > 0. 5 <u>and</u> plt > 50,000), whichever occurs first. If the marrow is hypocellular and without evidence of normal tri-lineage hematopoiesis the marrow should be repeated at Day 42

<sup>&</sup>lt;sup>4</sup> Follow-up for safety continues until the start of a new therapy (i.e. transplant preparative regimen) or Day 60 whichever occurs earlier (transplant related endpoints will be abstracted from the BMT database through the 1 year follow-up)

<sup>&</sup>lt;sup>5</sup> Intrathecal chemotherapy prophylaxis is allowed at the discretion of the treating physician.

<sup>&</sup>lt;sup>6</sup> Bone marrow must be sent for morphology, flow cytometry, standard cytogenetics, FISH and molecular testing for routine AML analysis.



#### 8. DRUG FORMULATION AND PROCUREMENT

8.1 Clofarabine

**8.1.1** Other Names: CLOLAR, clofarabine; CAFdA; Cl-F-ara-A

**8.1.2** Classification: Antineoplastic

- **8.1.3** Mode of Action: Clofarabine is sequentially metabolized intracellularly to the 5'monophosphate metabolite by deoxycytidine kinase and mono- and diphosphokinases to the active 5'-triphosphate metabolite. Clofarabine has high affinity for the activating phosphorylating enzyme, deoxycytidine kinase, equal to or greater than that of the natural substrate, deoxycytidine. Clofarabine inhibits DNA synthesis by decreasing cellular deoxynucleotide triphosphate pools through an inhibitory action on ribonucleotide reductase, and by terminating DNA chain elongation and inhibiting repair through incorporation into the DNA chain by competitive inhibition of DNA polymerases. The affinity of clofarabine triphosphate for these enzymes is similar to or greater than that of deoxyadenosine triphosphate. In preclinical models, clofarabine has demonstrated the ability to inhibit DNA repair by incorporation into the DNA chain during the repair process. Clofarabine 5'-triphosphate also disrupts the integrity of mitochondrial membrane, leading to the release of the pro-apoptotic mitochondrial proteins, cytochrome C and apoptosis-inducing factor, leading to programmed cell death. Clofarabine is cytotoxic to rapidly proliferating and quiescent cancer cell types in vitro. The population pharmacokinetics of clofarabine were studied in 40 pediatric patients aged 2 to 19 years (21 males/19 females) with relapsed or refractory ALL or AML. At the given 52 mg/m<sup>2</sup> dose, similar concentrations were obtained over a wide range of BSAs. Clofarabine was 47% bound to plasma proteins, predominantly to albumin. Based on non-compartmental analysis, systemic clearance and volume of distribution at steady-state were estimated to be 28.8 L/h/m<sup>2</sup> and 172 L/m<sup>2</sup>, respectively. The terminal half-life was estimated to be 5.2 hours. No apparent difference in pharmacokinetics was observed between patients with ALL and AML or between males and females. Based on 24-hour urine collections in the pediatric studies, 49-60% of the dose is excreted in the urine unchanged. In vitro studies using isolated human hepatocytes indicate very limited metabolism (0.2%), therefore the pathways of non-renal elimination remain unknown. Although no clinical drug-drug interaction studies have been conducted to date, on the basis of the *in vitro* studies, cytochrome p450 inhibitors and inducers are unlikely to affect the metabolism of clofarabine. The effect of clofarabine on the metabolism of cytochrome p450 substrates has not been studied. The pharmacokinetics of clofarabine have not been evaluated in patients with renal or hepatic dysfunction.
- **8.1.4** Storage and Stability: Clofarabine is a white to off-white solid with a melting point of 228°C to 230°C and a molecular weight of 303.5. The drug substance is very stable in the dry state, and aqueous solutions are stable to heat treatment.



Clofarabine is freely soluble in water (1.5 mg/mL) or buffered solutions at room temperature. Clofarabine is not less than 97% pure on a dried basis by high performance liquid chromatography (HPLC) analysis. Clofarabine is formulated at a concentration of 1 mg/mL. Clofarabine is supplied in 1 vial size: a 20-mL clear, glass vial with gray stopper and blue flip-off seal. The 20-mL vials contain 20 mL (20 mg) of sterile solution. The pH range of the solution is 4.5 to 7.5. The solution is clear and practically colorless, preservative free, and free from foreign matter. Store at 25°C (77°F); excursions permitted to 15-30°C (59-86°F).

Vials containing undiluted clofarabine for injection should be stored at controlled room temperature.

Store at 25°C (77°F); excursions permitted to 15-30°C (59-86°F). The commercial expiry period for clofarabine is 24 months at room temperature. Ongoing stability studies will continue to confirm the appropriate quality of drug product used for clinical trials beyond 24 months. Clofarabine for injection should be diluted with 0.9% sodium chloride injection USP or European Pharmacopeia (EP) normal saline (NS) or 5% dextrose injection (D5W) USP or EP prior to IV infusion. The resulting admixture may be stored at room temperature, but must be used within 24 hours of preparation.

- **8.1.5 Dose Specifics:** For the purposes of this study, clofarabine will be administered at the dose of 30 mg/m<sup>2</sup> for patients 0-30 years (20 mg/m<sup>2</sup> for patients > 30 years) IV over 2 hours (given at Hours 0 to 2) on Days 1 through 5.
- **8.1.6 Administration:** USP or 0.9% sodium chloride injection USP to a convenient volume such as the maximum final concentration should be between 0.15 mg/mL and 0.4 mg/mL, and infuse over 2 hours. The resulting admixture may be stored at room temperature, but must be used within 24 hours of preparation. To prevent drug incompatibilities, no other medications should be infused concurrently through the same IV lines as clofarabine. Also, no blood products should be administered at the same time as clofarabine.

To reduce the effects of tumor lysis and other adverse events it is recommended that continuous IV fluids be given throughout the 5 days of clofarabine administration. Since clofarabine is primarily excreted through the kidneys, drugs with known renal toxicity should be avoided during the 5 days of clofarabine administration. In addition, since the liver is a known target organ for clofarabine toxicity, concomitant use of medications known to induce hepatic toxicity should be avoided.

Pretreatment stress doses of steroids with hydrocortisone (50-100 mg/m<sup>2</sup>/dose IV daily) during clofarabine administration is allowed on this study.

- **8.1.7** Availability: Commercially available by prescription.
- **8.1.8** Side Effects: Refer to Appendix 4.

**Pregnancy Category D:** Clofarabine may cause fetal harm when administered to



a pregnant woman. Women of childbearing potential should be advised to avoid becoming pregnant while using Clofarabine. Men should be advised not to father a child while receiving treatment with Clofarabine, and for 2 months afterwards.

- 8.2 Cyclophosphamide
- **8.2.1 Other Names:** Cytoxan, CTX
- **8.2.2** Classification: Alkylating agent
- 8.2.3 Mode of Action: Cyclophosphamide is an alkylating agent related to nitrogen mustard. Cyclophosphamide is inactive until it is metabolized by P450 isoenzymes (CYP<sub>2</sub>B<sub>6</sub>, CYP<sub>2</sub>C<sub>9</sub>, and CYP<sub>3</sub>A<sub>4</sub>) in the liver to active compounds. The initial product is 4-hydroxycyclophosphamide (4-HC) which is in equilibrium with aldophosphamide which spontaneously releases acrolein to produce phosphoramide mustard. Phosphoramide mustard, which is an active bifunctional alkylating species, is 10 times more potent *in vitro* than is 4-HC and has been shown to produce interstrand DNA cross-link analogous to those produced by mechlorethamine. Approximately 70% of a dose of cyclophosphamide is excreted in the urine as the inactive carboxyphosphamide and 5-25% as unchanged drug. The plasma half-life ranges from 4.1 to 16 hours after IV administration.
- **8.2.4 Storage and Stability:** Cyclophosphamide for injection is available as powder for injection or lyophilized powder for injection in 500 mg, 1 g, and 2 g vials. The powder for injection contains 82 mg sodium bicarbonate/100 mg cyclophosphamide and the lyophilized powder for injection contains 75 mg mannitol/100 mg cyclophosphamide. Storage at or below 25°C (77°F) is recommended. The product will withstand brief exposures to temperatures up to 30°C (86°F).
- **8.2.5 Dose Specifics:** For the purposes of this study, cyclophosphamide 300 mg/m² will be administered intravenously over 30 to 60 minutes on Days 1 through 5.
- **8.2.6** Administration Cyclophosphamide for Injection: Reconstitute with Sterile Water or Bacteriostatic Water for Injection to a concentration of 20 mg/mL. Solutions reconstituted with preservative should be used within 24 hours if stored at room temperature or within 6 days if stored under refrigeration. If administered as undiluted drug at the 20 mg/mL concentration, reconstitute with NS only to avoid a hypotonic solution. Cyclophosphamide may be further diluted in dextrose or saline containing solutions for IV use.
- **8.2.7 Availability:** Cyclophosphamide is commercially available by prescription. Cyclophosphamide for Injection, USP contains cyclophosphamide monohydrate and is supplied in vials for single dose use.
- **8.2.8** Side Effects: Refer to Appendix 4.



**Pregnancy Category D:** Cyclophosphamide can cause fetal harm when administered to a pregnant woman.

- 8.3 Etoposide
- **8.3.1** Other Names: VP-16, Etopophos; Toposar; VePesid.
- **8.3.2** Classification: A semisynthetic derivative of podophyllotoxin that forms a complex with topoisomerase II and DNA which results in single and double strand DNA breaks. Its main effect appears to be in the S and G2 phase of the cell cycle. The initial t½ is 1.5 hours and the mean terminal half-life is 4 to 11 hours. It is primarily excreted in the urine. In children, approximately 55% of the dose is excreted in the urine as etoposide in 24 hours. The mean renal clearance of etoposide is 7 to 10 mL/min/m<sup>2</sup> or about 35% of the total body clearance over a dose range of 80 to 600 mg/m<sup>2</sup>. Etoposide, therefore, is cleared by both renal and non-renal processes, i.e., metabolism and biliary excretion. The effect of renal disease on plasma Etoposide clearance is not known. Biliary excretion appears to be a minor route of etoposide elimination. Only 6% or less of an intravenous dose is recovered in the bile as etoposide. Metabolism accounts for most of the non-renal clearance of etoposide. The maximum plasma concentration and area under the concentration time curve (AUC) exhibit a high degree of patient variability. Etoposide is highly bound to plasma proteins (~ 94%), primarily serum albumin. Pharmacodynamic studies have shown that etoposide systemic exposure is related to toxicity. Preliminary data suggests that systemic exposure for unbound etoposide correlates better than total (bound and unbound) etoposide. There is poor diffusion into the CSF < 5%. Cmax and AUC values for orally administered etoposide capsules consistently fall in the same range as the Cmax and AUC values for an intravenous dose of one-half the size of the oral dose. The overall mean value of oral capsule bioavailability is approximately 50% (range 25-75%). Etoposide phosphate is a water soluble ester of etoposide which is rapidly and completely converted to etoposide in plasma. Pharmacokinetic and pharmacodynamic data indicate that etoposide phosphate is bioequivalent to etoposide when it is administered in molar equivalent doses.
- **8.3.3 Dose Specifics:** For the purposes of this study, etoposide 100 mg/m<sup>2</sup> will be administered intravenously over 2 hours on Day 1 through 5.
- **8.3.4** Administration: Dilute etoposide to a final concentration ≤ 0.4 mg/mL in Dextrose or Normal Saline containing IV solutions. Etoposide infusions are stable at room temperature for 96 hours when diluted to concentrations of 0.2 mg/mL; stability is 24 hours at room temperature with concentrations of 0.4 mg/mL. The time to precipitation is highly unpredictable at concentrations > 0.4 mg/mL. Administer over 30 to 60 minutes; slow rate of administration if hypotension occurs. **Do not administer etoposide by rapid intravenous injection.** Use in-line filter during infusion secondary to precipitate formation risk. To avoid leaching of DEHP from PVC bags and tubing, prepare the etoposide solution as close as possible preferably within 4 hours to the time of administration or alternatively as per institutional policy, non-PVC containers and tubing may be used.



- **8.3.5** Availability: Commercially available by prescription.
- **8.3.6 Storage and Stability:** Etoposide for Injection is available in sterile multiple dose vials. The pH of the clear, nearly colorless to yellow liquid is 3 to 4. Each mL contains 20 mg etoposide, 2 mg citric acid, 30 mg benzyl alcohol, 80 mg modified polysorbate 80/tween 80, 650 mg polyethylene glycol 300, and 30.5 percent (v/v) alcohol. Vial headspace contains nitrogen. Unopened vials of etoposide are stable until expiration date on package at room temperature (25°C). Etoposide phosphate for injection is available for intravenous infusion as a sterile lyophilized powder in single-dose vials containing etoposide phosphate equivalent to 100 mg etoposide, 32.7 mg sodium citrate *USP*, and 300 mg dextran 40. Etoposide phosphate must be stored under refrigeration 2°-8°C (36°-46°F). Unopened vials of Etoposide phosphate are stable until the expiration date on the package.
- **8.3.7 Side Effects:** Refer to Appendix 4.

**Pregnancy Category D:** Etoposide may cause fetal harm when administered to a pregnant woman. Women of childbearing potential should be advised to avoid becoming pregnant while using Etoposide. Men should be advised not to father a child while receiving treatment with Etoposide, and for 2 months afterwards.

# 9. ADVERSE EVENT MONITORING, DOCUMENTATION, AND REPORTING

Toxicity and adverse events will be classified according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE) and reported on the schedule below. A copy of the CTCAE can be downloaded from the CTEP home page: <a href="http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40">http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40</a>

#### 9.1 **Definitions**

The following definitions are based on the Code of Federal Regulations Title 21 Part 312.32 (21 CFR 312.32(a)).

**Adverse Event:** Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

**Suspected Adverse Reaction:** Any adverse event for which there is a reasonable possibility that the drug caused the adverse event.

**Life-Threatening Adverse Event Or Life-Threatening Suspected Adverse Reaction:** An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death.

**Event Attribution Categories:** CTCAE does not define an AE as necessarily 'caused by a therapeutic intervention.' The clinical investigator must assign attribution for an adverse



event after naming and grading of the event.

| Attribution | Description |
|-------------|---------------------------------------------------|
| Unrelated | The AE is clearly NOT related to the intervention |
| Unlikely | The AE is doubtfully related to the intervention |
| Possible | The AE may be related to the intervention |
| Probable | The AE is likely related to the intervention |
| Definite | The AE is clearly related to the intervention |

Unanticipated (unexpected) adverse event or unexpected suspected adverse reaction as defined by the Medical College of Wisconsin IRB are those that are *not* already described as potential risks in the consent form, *not* listed in the Investigator's Brochure or *not* part of an underlying disease.

**Expedited (Rapid) Reporting:** Certain events may require rapid notification to entities providing patient safety oversight (i.e. IRB) as detailed in Section 9.3.

#### 9.2 Adverse Event Documentation

Adverse events occurring after the initiation of any study treatment must be documented. Refer to Appendix 4 for a list of expected toxicities.

Since a key endpoint of this study is to characterize the toxicities of clofarabine, cyclophosphamide and etoposide when used in combination, adverse event documentation requirements will be determined based on grade, expectedness and relationship to study therapy as follows:

| | Grade 1 | Grade 2 | | Grade 3 | | Grade 4 and 5 |
|---|---|---|---|---|---|---|
| | Expected or | Expected | Unexpected | Expected | Unexpected | Expected or |
| | Unexpected | | | | | Unexpected |
| Unrelated | Not required | Not | Not required | Not | Required | Required |
| Unlikely | | required | | Required | | |
| Possible | Not required | Not | Not Required | Not | Required | Required |
| Probable | | required | | Required | (Non | |
| Definite | | | | | hematologic only) | |

**Stopping Rule Events:** The following events count toward a study stopping rule per Section 11.4 and must be reported to the MCW Study Coordinator and Dr. Burke using the SAE Form found in REDCap which is also immediately reported (within 24 hours of PI notification) to the MCW DSMC:

- Any Grade 4 non-hematologic treatment related event
- Any death, regardless of cause during the reporting period for this study (from initiation of study treatment through the start of a new treatment (i.e. transplant preparative regimen), or Day 60, whichever occurs earlier)



All patients will be monitored until the start of a new treatment (i.e. transplant preparative regimen) or Day 60, whichever occurs earlier, as it is expected that most treatment related adverse events will occur during this period.

For patients who go on to transplant, transplant related endpoints will be collected by record review.

# 9.3 Adverse Event Reporting Requirements

The reporting period for this study is from initiation of study treatment through the start of a new treatment (i.e. transplant preparative regimen), or D ay 60, whichever occurs earlier; however after this time point, the investigator must report upon knowledge any study treatment related event meeting the <u>expedited</u> reporting criteria listed in the following table.

| Agency | Criteria for Reporting | Timeframe | Form to | Copy AE |
|---|---|---|---|---|
| | | | Use | To: |
| MCW<br>IRB | UPIRSO: Any event which is unanticipated, involved new or increased risk to subjects, and was at least possibly related to study procedures through Day 60 or the start of a new treatment whichever is earlier Other Problems or Events meeting the | 5 calendar<br>days after<br>PI<br>Notification | SAE Found<br>in REDCap | Dr. Michael<br>Burke &<br>MCW Study<br>Coordinator |
| MCW<br>DSMC | definition of UPIRSO Any event that counts toward a study stopping rule (see Section 11.4) | Within 24<br>hours of PI<br>notification | SAE Found<br>in REDCap | Dr. Michael<br>Burke &<br>MCW Study<br>Coordinator |

Serious adverse events are reported directly to Dr. Michael Burke and the MCW Study Coordinator within 72 hours of the event via the REDCap database (Section 10.1). The adverse event report is reviewed by Dr. Michael Burke and Causality/Attribution assigned, as applicable.

MCW CC DSMC Reporting: The MCW Cancer Center DSMC is responsible for the global oversight and review of patient safety on this clinical trial. The DSMC meets twice a year (at a minimum) and all submitted outcome data is reviewed including all adverse events reported to the MCW IRB. The DSMC reserves the right to meet more frequently on an as needed basis based on the events submitted.

The DSMC semi-annual review confirms that the trial has not met any stopping rules and reviews any patient safety problems necessitating discontinuation of the trial. A report from the DSMC is submitted to the MCW IRB as well as the trial coordinators/local PIs of this protocol.

Grade 3 Unexpected (non-hematological only), and all Grade 4 and 5 events will be submitted to the DSMC within 24 hours of PI (Dr. Michael Burke) Notification. The DSMC will acknowledge the submission with a responding email.



MCW IRB Reporting: Serious adverse events are reported directly to the PI and the MCW Study Coordinator within 72 hours of the event via the REDCap database (Section 10.1). The adverse event report is reviewed by Dr. Michael Burke and Causality/Attribution assigned, as applicable. If the adverse event meets the MCW IRB criteria for expedited reporting, an official signed report is submitted to the MCW Institutional Review Board. All deaths, regardless of the cause, are reported to the MCW IRB.

An official report of a serious adverse event is faxed or emailed to the MARCH coordinating center within five days of occurrence.

## 9.4 Event Notification, Deviations, or Patient Complaints

Any event, protocol deviation, or patient complaint, not meeting the criteria for serious adverse event reporting, should be reported to the MCW Study Coordinator via the REDCap database (Section 10.1). The report is reviewed by the PI and any further action, if deemed necessary, is discussed with the reporting site.

#### 10. STUDY DATA COLLECTION AND MONITORING

## 10.1 Data Management

Data management will be performed utilizing an electronic data capture system called REDCap. REDCap (Research Electronic Data Capture) is a secure, web-based application designed exclusively to support data capture for research studies.

Security is provided through a table based authentication system where users are added to a project and are granted specific rights within the project(s) they have access to. These specific access rights consist of access to the study calendar, 3 levels (no access, deidentified, full data set) of access to the Data Export Tool, access to the Data Import Tool, the Data Comparison tool (used when double-data entry is utilized), access to the complete logging records, the File Repository, User Rights (ability to add users and grant rights), access Data Access Groups, access to reports and the report builder, access for project setup and design, and a few more. Users can only access the specific projects they have been granted access to.

The CTSI of Southeast Wisconsin's REDCap installation is housed on a CTSI-owned server located in the TBRC Data Center at the Medical College of Wisconsin, and all traffic between the user's browser and the server is encrypted with a 128-bit Digicert SSL certificate. The server OS is incrementally backed up nightly and rotated off-site. The database (MySQL) is backed up 4 times daily and is also part of the incremental nightly OS back up.

The Data Access Groups feature within REDCap will be enabled for this project. This feature allows users to be designated into groups (sites), after which any user in the Data Access Group may only see records created by another person in that group. Thus, sites may enter patient data but not be allowed to see other site's data/records. Only the CDCC will be able to view and analyze data entered from all site records. The data export function is included as part of the website. Once data has been successfully entered into



the database, the investigator and his/her staff can extract this data for different analysis software programs.

Once an institution consents a patient, they will enter the patient demographics into the REDCap system which will assign a study ID. Centers will be required to upload the signed informed consent to the CDCC office via the REDCap database. Subsequent data will be entered via REDCap for review by the CDCC in the same manner. The study coordinator will review the data reports with Dr. Burke within 24-72 hours The overall study coordinator will follow-up with the institution if there are missing or delinquent data forms, and request submission within a timely manner.

Any paper data (i.e. safety reports, reports generated from REDCap) will be kept in a locked and secure location within the Clinical Trials Office of the Pediatric Hematology/Oncology and Bone Marrow Transplant Program. The Clinical Trials Office has secure, electronic employee badge access only. Any paper data that is generated and pertinent to the conduct of study, will be kept for 10 years after the study file is closed with the IRB.

REDCap training will be provided by the MCW Clinical and Translational Science Institute (CTSI) to each participating site.

For patients going on to transplant, the transplant related endpoints for this study will be collected by record review for 3 years post-transplant.

# **10.2** Case Report Forms

**Initial Plans:** Participant data will be collected using protocol specific case report forms developed by the MACC Fund Center CTO. The CRFs will be approved by the study's Principal Investigator and the Biostatistician prior to release for use. The Study Coordinator or designee will be responsible for registering the patient at time of study entry, completing CRFs based on the patient specific calendar or roadmap, and updating the patient record until the end of required study participation.

**Implementation of REDCap:** Participant data will be collected using protocol specific electronic case report forms (e-CRFs) developed within REDCap based on its library of standardized forms. The e-CRF will be approved by the study's Principal Investigator and the Biostatistician prior to release for use. The Study Coordinator or designee will be responsible for registering the patient into REDCap at time of study entry, completing e-CRFs based on the patient specific calendar, and updating the patient record until the end of required study participation.

#### 10.3 Data and Safety Monitoring Plan (DSMP)

The study's Data and Safety Monitoring Plan will be in compliance with the Medical College of Wisconsin Cancer Center's Data & Safety Monitoring Plan (DSMP), which can be accessed at <a href="http://www.mcw.edu/FileLibrary/Groups/HumanResearchProtectionOffice/IRB/Newandown-nd-braftPolicies/IRBSOPDSMP.pdf">http://www.mcw.edu/FileLibrary/Groups/HumanResearchProtectionOffice/IRB/Newandown-nd-braftPolicies/IRBSOPDSMP.pdf</a>



This study will be reviewed by the Medical College of Wisconsin Cancer Center Data Safety Monitoring Committee (MCW CC DSMC). A summary of the MCW CC DSMC activities are as follows:

- Review the clinical trial for data integrity and safety
- Review all Grade 3 unexpected adverse events, all Grade 4 and 5 adverse events, and all events requiring expedited reporting as defined per protocol
- Review all DSM reports
- Submit a summary of any recommendations related to study conduct
- Terminate the study if deemed unsafe for patients

A copy of the MCW CC Data and Safety Monitoring Plan and membership roster will be maintained in the study research file and updated as membership changes. The committee will review reports from the study PI twice annually (or more frequently if needed) and provide recommendations on trial continuation, suspension or termination as necessary.

Any available DSMC letters will be submitted to the IRB of record as required.

For the purposes of data and safety monitoring, this study is classified as moderate risk. Therefore the following requirements will be fulfilled:

- The PI will complete and submit a semi-annual Trial Progress Report to the MCW Cancer Center Data and Safety Monitoring Committee (DSMC) with the understanding the MCW DSMC may require more frequent reporting.
- The PI will oversee the submission of all reportable events per the definition of reportable in Section 9.3 to the MCW Cancer Center's DSMC and the MCW IRB.

### 10.4 Monitoring

The PI at each participating center is responsible for monitoring this study for accuracy of data and protocol compliance at their institution. Patient eligibility will be confirmed by Dr. Michael Burke before each patient is enrolled.

The PI, data coordinators, and research nurses are responsible for review and maintenance of all patient records at their individual institution to ensure data integrity and protocol adherence.

The site PI will permit study-related monitoring, audits, and inspections by the MCW compliance groups, as necessary. The investigator will make available all study related documents (i.e. source documents, regulatory documents, data collection instruments, study data, etc.). The investigator will ensure the capability for inspections of applicable study-related facilities (i.e. pharmacy, diagnostic laboratory, etc.) will be available for trial related monitoring, audits, or regulatory inspections.

#### 10.5 Record Retention

The investigator will retain study records including source data, copies of case report forms, consent forms, HIPAA authorizations, and all study correspondence in a secured


facility for 10 years after the study file is closed with the IRB.

In addition, the Clinical Trials Office (CTO) will keep a master log of all patients participating in the study with sufficient information to allow retrieval of the medical records for that patient. Please contact the CTO before destroying any study related records.

### 11. STATISTICAL CONSIDERATIONS

This is a Phase 2 study designed for the purpose of estimating the key parameters for use in future studies and for estimating whether there is a difference between adult and pediatric response.

### 11.1 Statistic Endpoints

The following parameters will be monitored and used to estimate the effect sizes with their 95% confidence intervals.

- The effect of Clofarabine, Cyclophosphamide, and Etoposide in eliminating the presence of persistent disease without causing a significant delay of HCT due to treatment related toxicity, defined as greater than 56 days from completion of bridging therapy to start of HCT. The proportion of any toxicities associated with Clofarabine, Cyclophosphamide, and Etoposide
- The proportion of pre-transplant chemotherapy-induced aplasia (defined as greater than 42 days after infusion of chemotherapy)
- The proportion of infectious complications following bridging therapy and before HCT
- The proportion of patients who do not proceed to HCT after receiving bridging therapy due to disease status or treatment related morbidity/mortality
- Treatment-related mortality at Day 100 after HCT
- One year disease-free survival after HCT
- One year overall survival after HCT
- The proportion of relapse within one year of HCT

### 11.2 Statistical Analysis

SAS 9.4 (Cary, NC, USA) will be used for the statistical analyses. The summary statistics including 95% confidence intervals for MRD negative conversion rate will be calculated. All toxicity and safety assessments will be presented in the data listings and summarized with point estimates and 95% confidence intervals. Proportions will use exact binomial confidence intervals. Overall survival and disease free survival estimates after HCT will use the Kaplan-Meier method. The Nelson-Aalen counting process method will be used to estimate cumulative survival/relapse and the intensity of the process. Relapse and treatment-related mortality after HCT will be estimated by competing risk analysis using the counting process approach.

### 11.3 Sample Size Justification

This is a Phase 2 study designed for the purpose of estimating the following key



parameters for use in future studies and for estimating whether there is a difference between young adult and pediatric response: 1) The effect of CCE in eliminating the presence of MRD; 2) Whether CCE will significantly delay time to HCT due to treatment related toxicity; 3) The proportion of any toxicities associated with CCE; 4) The proportion of pre-transplant chemotherapy-induced aplasia (defined as greater than 42 days after infusion of chemotherapy); 5) The proportion of infectious complications following bridging therapy and before HCT; 6) The proportion of patients who do not proceed to HCT after receiving bridging therapy due to disease status or treatment related morbidity/mortality; 7) Treatment—related mortality at Day 100 after HCT; 6) One year DFS after HCT; 7) One year OS after HCT; and 8) The proportion of relapse within 1-year of HCT. Post-HCT outcomes (OS, EFS and Relapse) will be compared to historical controls for children, adolescent and young adults (separated by age; 0-18 and 19-39 years) receiving a HCT for ALL or AML with pre-HCT MRD, using national and international data.

### 11.4 Early Stopping Rule for Excessive Toxicity (pre-HCT) and TRM (post-HCT)

The complications and adverse events will be closely monitored in this study. Rates of grade 3 or greater non hematologic toxicity that does not resolve by day 56 following bridging therapy, such that patients are not able to proceed to HCT on time, that exceed 10% will be considered unacceptable. The trial will be stopped for review if the Grade 3 non-hematologic toxicity rate statistically exceeds 10%. Similarly, a pre-HCT toxic death rate attributed to the bridging therapy that exceeds p0=5% will be considered unacceptable. No formal statistical rule will be employed. Rather, if the crude proportion of patients experiencing a toxic death exceed 5% at any time (using the Kaplan-Meier curve and log-rank comparisons) prior to HCT, the cause and circumstances of these deaths will be reviewed with the study committee and with the Data and Safety Monitoring Committee to determine whether modifications to or termination of the study is warranted. As well, if we see a lack of efficacy in the ability of this regimen to eliminate MRD at 1/3 or 2/3 the total number of patients, the study will be suspended to consider dose escalation of clofarabine.

| Nth<br>Patient | Stopping<br>Number<br>Mortality | Stopping<br>Number<br>Toxicity | Nth<br>Patient | Stopping<br>Number<br>Mortality | Stopping<br>Number<br>Toxicity |
|---|---|---|---|---|---|
| 1 | - | - | 14 | 3 | 4 |
| 2 | - | - | 15 | 3 | 5 |
| 3 | 2 | 2 | 16 | 3 | 5 |
| 4 | 2 | 2 | 17 | 4 | 5 |
| 5 | 2 | 3 | 18 | 4 | 5 |
| 6 | 2 | 3 | 19 | 4 | 5 |
| 7 | 2 | 3 | 20 | 4 | 6 |
| 8 | 3 | 3 | 21 | 4 | 6 |
| 9 | 3 | 3 | 22 | 4 | 6 |
| 10 | 3 | 4 | 23 | 4 | 6 |
| 11 | 3 | 4 | 24 | 4 | 6 |



| 12 | 3 | 4 | 25 | 4 | 7 |
|----|---|---|----|---|---|
| 13 | 3 | 4 | | | |

#### 12. CONDUCT OF THE STUDY

#### 12.1 Good Clinical Practice

The study will he conducted in accordance with appropriate the regulatory requirement(s). The investigator will be thoroughly familiar with the appropriate use of the drug as described in the protocol and Investigator's Brochure. Essential clinical documents will be maintained to demonstrate the validity of the study and the integrity of the data collected. Master files should be established at the beginning of the study, maintained for the duration of the study and retained according to the appropriate regulations.

### 12.2 Ethical Considerations

The study will be conducted in accordance with ethical principles founded in the Declaration of Helsinki. The IRB will review all appropriate study documentation in order to safeguard the rights, safety and well-being of the patients. The study will only be conducted at sites where IRB approval has been obtained. The protocol, informed consent, written information given to the patients, safety updates, annual progress reports, and any revisions to these documents will be provided to the IRB by the investigator.

#### 12.3 Informed Consent

All potential study participants will be given a copy of the MCW IRB approved consent to review. The investigator or designee will explain all aspects of the study in lay language and answer all questions regarding the study. If the participant (or parents/guardians for a minor) decides to participate in the study, he/she will be asked to sign and date the consent document. Patients who refuse to participate or who withdraw from the study will be treated without prejudice.

### 12.4 Clinical Trial Registration

A description of this clinical trial will be available at: <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time. NCI Number: NCT02349178



### **REFERENCES**

- 1. Miglino M, Berisso G, Grasso R, Canepa L, Clavio M, Pierri I *et al.* Allogeneic bone marrow transplantation (BMT) for adults with acute lymphoblastic leukemia (ALL): predictive role of minimal residual disease monitoring on relapse. *Bone marrow transplantation* 2002; 30(9): 579-585. doi: 10.1038/sj.bmt.1703659
- 2. Knechtli CJ, Goulden NJ, Hancock JP, Grandage VL, Harris EL, Garland RJ *et al.* Minimal residual disease status before allogeneic bone marrow transplantation is an important determinant of successful outcome for children and adolescents with acute lymphoblastic leukemia. *Blood* 1998; 92(11): 4072-4079.
- 3. Foster JH, Hawkins DS, Loken MR, Wells DA, Thomson B. Minimal residual disease detected prior to hematopoietic cell transplantation. *Pediatric blood & cancer* 2011; 57(1): 163-165. doi: 10.1002/pbc.23079
- 4. Venditti A, Maurillo L, Buccisano F, Del Poeta G, Mazzone C, Tamburini A *et al.* Pretransplant minimal residual disease level predicts clinical outcome in patients with acute myeloid leukemia receiving high-dose chemotherapy and autologous stem cell transplantation. *Leukemia* 2003; 17(11): 2178-2182. doi: 10.1038/sj.leu.2403138
- 5. Wertheim GB, Bagg A. Minimal residual disease testing to predict relapse following transplant for AML and high-grade myelodysplastic syndromes. *Expert review of molecular diagnostics* 2011; 11(4): 361-366. doi: 10.1586/erm.11.19
- 6. Jacobsohn DA, Tse WT, Chaleff S, Rademaker A, Duerst R, Olszewski M *et al.* High WT1 gene expression before haematopoietic stem cell transplant in children with acute myeloid leukaemia predicts poor event-free survival. *British journal of haematology* 2009; 146(6): 669-674. doi: 10.1111/j.1365-2141.2009.07770.x
- 7. Bader P, Kreyenberg H, Henze GH, Eckert C, Reising M, Willasch A *et al.* Prognostic value of minimal residual disease quantification before allogeneic stem-cell transplantation in relapsed childhood acute lymphoblastic leukemia: the ALL-REZ BFM Study Group. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2009; 27(3): 377-384. doi: 10.1200/JCO.2008.17.6065
- 8. Pulsipher MA, Bader P, Klingebiel T, Cooper LJ. Allogeneic transplantation for pediatric acute lymphoblastic leukemia: the emerging role of peritransplantation minimal residual disease/chimerism monitoring and novel chemotherapeutic, molecular, and immune approaches aimed at preventing relapse. *Biology of blood and marrow transplantation: journal of the American Society for Blood and Marrow Transplantation* 2009; 15(1 Suppl): 62-71. doi: 10.1016/j.bbmt.2008.11.009
- 9. Goulden N, Bader P, Van Der Velden V, Moppett J, Schilham M, Masden HO *et al.* Minimal residual disease prior to stem cell transplant for childhood acute lymphoblastic



leukaemia. British journal of haematology 2003; 122(1): 24-29.

- 10. Krejci O, van der Velden VH, Bader P, Kreyenberg H, Goulden N, Hancock J *et al.* Level of minimal residual disease prior to haematopoietic stem cell transplantation predicts prognosis in paediatric patients with acute lymphoblastic leukaemia: a report of the Pre-BMT MRD Study Group. *Bone marrow transplantation* 2003; 32(8): 849-851. doi: 10.1038/sj.bmt.1704241
- 11. Sramkova L, Muzikova K, Fronkova E, Krejci O, Sedlacek P, Formankova R *et al.* Detectable minimal residual disease before allogeneic hematopoietic stem cell transplantation predicts extremely poor prognosis in children with acute lymphoblastic leukemia. *Pediatric blood & cancer* 2007; 48(1): 93-100. doi: 10.1002/pbc.20794
- 12. Society AC. Cancer Facts and Figures. American Cancer Society 2007; Atlanta, GA.
- 13. Walter RB, Gooley TA, Wood BL, Milano F, Fang M, Sorror ML *et al.* Impact of pretransplantation minimal residual disease, as detected by multiparametric flow cytometry, on outcome of myeloablative hematopoietic cell transplantation for acute myeloid leukemia. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2011; 29(9): 1190-1197. doi: 10.1200/JCO.2010.31.8121
- 14. Walter RB, Buckley SA, Pagel JM, Wood BL, Storer BE, Sandmaier BM *et al.* Significance of minimal residual disease before myeloablative allogeneic hematopoietic cell transplantation for AML in first and second complete remission. *Blood* 2013; **122**(10): 1813-1821. doi: 10.1182/blood-2013-06-506725
- 15. Valkova V, Polak J, Markova M, Vitek A, Hajkova H, Salek C *et al.* Minimal residual disease detectable by quantitative assessment of WT1 gene before allogeneic stem cell transplantation in patients in first remission of acute myeloid leukemia has an impact on their future prognosis. *Clin Transplant* 2013; 27(1): E21-29. e-pub ahead of print 2012/12/13; doi: 10.1111/ctr.12046
- 16. Wang Y, Liu DH, Liu KY, Xu LP, Zhang XH, Han W *et al.* Impact of pretransplantation risk factors on post transplantation outcome of patients with acute myeloid leukemia in remission after haploidentical hematopoietic stem cell transplantation. *Biol Blood Marrow Transplant* 2013; 19(2): 283-290. e-pub ahead of print 2012/10/16; doi: 10.1016/j.bbmt.2012.10.002
- 17. Schnittger S, Kern W, Tschulik C, Weiss T, Dicker F, Falini B *et al.* Minimal residual disease levels assessed by NPM1 mutation-specific RQ-PCR provide important prognostic information in AML. *Blood* 2009; 114(11): 2220-2231. doi: 10.1182/blood-2009-03-213389
- 18. Kwon M, Martinez-Laperche C, Infante M, Carretero F, Balsalobre P, Serrano D *et al.* Evaluation of minimal residual disease by real-time quantitative PCR of Wilms' tumor 1 expression in patients with acute myelogenous leukemia after allogeneic stem cell transplantation: correlation with flow cytometry and chimerism. *Biology of blood and marrow transplantation: journal of the American Society for Blood and Marrow*



Transplantation 2012; 18(8): 1235-1242. doi: 10.1016/j.bbmt.2012.01.012

- 19. Oran B, Singleton T, Ramirez PA, Shanley R, Brunstein C, Ustun C *et al.* Allogeneic Hematopoietic Stem Cell Transplantation Overcomes the Adverse Prognostic Impact of Minimal Residual Disease in Acute Myeloid Leukemia. *ASH Annual Meeting Abstracts* 2011; 118(21): 2027-.
- 20. Bachanova V, Burke MJ, Yohe S, Cao Q, Sandhu K, Singleton TP *et al.* Unrelated cord blood transplantation in adult and pediatric acute lymphoblastic leukemia: effect of minimal residual disease on relapse and survival. *Biology of blood and marrow transplantation: journal of the American Society for Blood and Marrow Transplantation* 2012; 18(6): 963-968. doi: 10.1016/j.bbmt.2012.02.012
- 21. Raetz EA, Borowitz MJ, Devidas M, Linda SB, Hunger SP, Winick NJ *et al.* Reinduction platform for children with first marrow relapse of acute lymphoblastic Leukemia: A Children's Oncology Group Study[corrected]. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2008; 26(24): 3971-3978. doi: 10.1200/JCO.2008.16.1414
- 22. Dreyer ZE, Dinndorf PA, Camitta B, Sather H, La MK, Devidas M *et al.* Analysis of the role of hematopoietic stem-cell transplantation in infants with acute lymphoblastic leukemia in first remission and MLL gene rearrangements: a report from the Children's Oncology Group. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2011; 29(2): 214-222. doi: 10.1200/JCO.2009.26.8938
- 23. Trifilio S, Zhou Z, Altman J, Frankfurt O, Pantiru M, Mehta J. Dose-intense etoposide-cyclophosphamide without stem cell transplantation for patients with intermediate and high cytogenetic risk primary refractory and relapsed acute myeloid leukemia. *Leukemia research* 2013; 37(8): 872-876. doi: 10.1016/j.leukres.2013.05.006
- 24. Miano M, Pistorio A, Putti MC, Dufour C, Messina C, Barisone E *et al.* Clofarabine, cyclophosphamide and etoposide for the treatment of relapsed or resistant acute leukemia in pediatric patients. *Leukemia & lymphoma* 2012; 53(9): 1693-1698. doi: 10.3109/10428194.2012.663915
- 25. Hijiya N, Thomson B, Isakoff MS, Silverman LB, Steinherz PG, Borowitz MJ *et al.* Phase 2 trial of clofarabine in combination with etoposide and cyclophosphamide in pediatric patients with refractory or relapsed acute lymphoblastic leukemia. *Blood* 2011; 118(23): 6043-6049. doi: 10.1182/blood-2011-08-374710
- 26. Clofarabine Investigator's Brochure. 6th ed. San Antonio, TX: Genzyme Corp. 2007.
- 27. Jeha S, Gandhi V, Chan KW, McDonald L, Ramirez I, Madden R *et al.* Clofarabine, a novel nucleoside analog, is active in pediatric patients with advanced leukemia. *Blood* 2004; 103(3): 784-789. doi: 10.1182/blood-2003-06-2122
- 28. Lotfi K, Mansson E, Spasokoukotskaja T, Pettersson B, Liliemark J, Peterson C *et al.* Biochemical pharmacology and resistance to 2-chloro-2'-arabino-fluoro-2'-deoxyadenosine, a novel analogue of cladribine in human leukemic cells. *Clinical cancer*



- research: an official journal of the American Association for Cancer Research 1999; 5(9): 2438-2444.
- 29. Jeha S, Gaynon PS, Razzouk BI, Franklin J, Kadota R, Shen V *et al.* Phase II study of clofarabine in pediatric patients with refractory or relapsed acute lymphoblastic leukemia. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2006; 24(12): 1917-1923. doi: 10.1200/JCO.2005.03.8554
- 30. Burnett AK, Russell NH, Kell J, Dennis M, Milligan D, Paolini S *et al.* European development of clofarabine as treatment for older patients with acute myeloid leukemia considered unsuitable for intensive chemotherapy. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2010; 28(14): 2389-2395. doi: 10.1200/JCO.2009.26.4242
- 31. Faderl S, Ravandi F, Huang X, Wang X, Jabbour E, Garcia-Manero G *et al.* Clofarabine plus low-dose cytarabine followed by clofarabine plus low-dose cytarabine alternating with decitabine in acute myeloid leukemia frontline therapy for older patients. *Cancer* 2012; 118(18): 4471-4477. doi: 10.1002/cncr.27429
- 32. Jeha S, Razzouk B, Rytting M, Rheingold S, Albano E, Kadota R *et al.* Phase II study of clofarabine in pediatric patients with refractory or relapsed acute myeloid leukemia. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2009; 27(26): 4392-4397. doi: 10.1200/JCO.2008.18.8706
- 33. Styczynski J, Gil L, Derwich K, Wachowiak J, Balwierz W, Badowska W *et al.* Comparison of clofarabine activity in childhood and adult acute leukemia: individual tumor response study. *Anticancer research* 2009; 29(5): 1643-1650.
- 34. Karp JE, Ricklis RM, Balakrishnan K, Briel J, Greer J, Gore SD *et al.* A Phase 1 clinical-laboratory study of clofarabine followed by cyclophosphamide for adults with refractory acute leukemias. *Blood* 2007; 110(6): 1762-1769. doi: 10.1182/blood-2007-03-081364
- 35. Kantarjian HM, Erba HP, Claxton D, Arellano M, Lyons RM, Kovascovics T *et al.* Phase II study of clofarabine monotherapy in previously untreated older adults with acute myeloid leukemia and unfavorable prognostic factors. *Journal of clinical oncology: official journal of the American Society of Clinical Oncology* 2010; 28(4): 549-555. doi: 10.1200/JCO.2009.23.3130
- 36. Foster MC, Amin C, Voorhees PM, van Deventer HW, Richards KL, Ivanova A *et al.* A Phase I dose- escalation study of clofarabine in combination with fractionated gemtuzumab ozogamicin in patients with refractory or relapsed acute myeloid leukemia. *Leukemia & lymphoma* 2012; 53(7): 1331-1337. doi: 10.3109/10428194.2011.647313
- 37. Amadori S, Stasi R, Martelli AM, Venditti A, Meloni G, Pane F *et al.* Temsirolimus, an mTOR inhibitor, in combination with lower-dose clofarabine as salvage therapy for older patients with acute myeloid leukaemia: results of a phase II GIMEMA study (AML-1107). *British journal of haematology* 2012; 156(2): 205-212. doi: 10.1111/j.1365-2141.2011.08940.x



- 38. Gossai N, Verneris MR, Karras NA, Gorman MF, Patel NJ, Burke MJ. A clofarabine-based bridging regimen in patients with relapsed ALL and persistent minimal residual disease (MRD). *Bone marrow transplantation* 2013. doi: 10.1038/bmt.2013.195
- 39. Tischer J, Stemmler HJ, Engel N, Hubmann M, Fritsch S, Prevalsek D *et al.* Feasibility of clofarabine cytoreduction followed by haploidentical hematopoietic stem cell transplantation in patients with relapsed or refractory advanced acute leukemia. *Annals of hematology* 2013; 92(10): 1379-1388. doi: 10.1007/s00277-013-1862-6



### APPENDIX 1 Eligibility Checklist

| | Eligibil | lity Checklist - | - Page 1 of 2 | | | | |
|---|---|---|---|---|---|---|---|
| | _ | Initials | | | Patient ID | | |
| | Date Co | onsent Form Si | igned://_ | Dia | agnosis ALL or AML | | |
| | Inclusion | on Criteria | | | | | |
| | A "NO" | " response to a | ny of the following disqua | alifies the patien | nt from study entry. | | |
| | | | | | | Yes | No |
| 1 | Diagnosis of | acute lymphobla | stic leukemia (ALL) or acute | myeloid leukemis | a (AML) with < 5% blasts in the | | |
| | | | logy and that meets the follow | | a (711112) with 570 blasts in the | | |
| | | | of PD ( $\geq 0.01\%$ leukemic blast | • | 5% leukemic blasts for AML | | |
| | | e bone marrow) | (= | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | |
| | OR | , | | | | | |
| | Molecular Molecular | r/cytogenetic evid | lence of disease (FISH or PCR | methodology) per | formed within 7 days and with the | | |
| | | | neic hematopoietic cell transpl | | | | |
| 2 | Age 0 to 39 y | | | | | | |
| 3 | Karnofsky ≥ :<br>Score - □□ | 50% for patients □ | 16 years and older and Lansky | status $\geq 50$ for pat | ients under 16 years of age | | |
| 4<br>5 | | | | | | | |
| 5 | Adequate org | an function define | ed as within 7 days of the start | of study treatment, | unless otherwise noted | | |
| | | T | | | | | |
| | Test | R | Required Value | Patient's Resi | ult Date Performed | | |
| | Creatinine | | ance $\geq 60 \text{ mL/min/1.73m}^2$ | | | | |
| | | OR serum creat | inine based on age: | mL/min/1.73 m <sup>2</sup> | | | |
| | | Age (Yrs) | Maximum Serum | OR | | | |
| | | 1190 (110) | Creatinine (mg/dl) | OK | | | |
| | | 2 to < 6 | 0.8 0.8 | . mg/dl | | | |
| | | 6 to < 10 | 1.0 1.0 | | | | |
| | | 10 to < 13 | 1.2 1.2 | | | | |
| | | 13 to < 16 | 1.5 1.4 | | | | |
| | | ≥ 16 | 1.7 1.4 | | | | |
| | Total<br>Bilirubin | $\leq$ 1.5 x ULN for | age | | | | |
| | ALT | < 5 X ULN | | | | | |
| | Cardiac | Left ventricular<br>ECHO/MUGA | ejection fraction ≥ 40% by | % | | | |
| 6 | Patients must | | ered from the acute toxic effec | ts of all prior chem | notherapy, immunotherapy, or | | |
| Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. At least 7 days must have elapsed from prior chemotherapy. | | | | | | | |
| | | | | oletion of therapy v | with a growth factor and at least 14 | | |
| days since pegfilgrastim (Neulasta®) administration. | | | | | | | |
| 7 | | | | | ontraception (diaphragm, birth | | |
| | | | | | aneous implants, or abstinence, | | |
| | | | ent and for 2 months after the | | | | |
| | _ | | aceptive for the duration of tre | aunent and for 2 m | ionuis after the fast dose of | | |
| chemotherapy. | | | | | | | |



| 8 | Voluntary written consent before performance of any study-related procedure not part of normal medical care, |
|---|---|
| | with the understanding that consent may be withdrawn by the subject/guardian at any time without prejudice to |
| | future medical care. |

| | APPENDIX I Eligibility Checklist - Continued | | |
|---|---|---|---|
| | Eligibility Checklist – Page 2 of 2 Patient Initials | | |
| | Exclusion Criteria | | |
| | A "Yes" response to any of the following disqualifies the patient from study entry. | <b>T T</b> 7 | l ».r |
| _ | | Yes | No |
| 9 | Acute Promyelocytic Leukemia (APL) | | |
| 10 | Active CNS leukemia or presence of chloromatous disease | <u> </u> | |
| 11 | Receiving concomitant chemotherapy, radiation therapy; immunotherapy or other anti-cancer therapy other than | | |
| 10 | is specified in the protocol | <u> </u> | - |
| 12 | Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms | | |
| 13 | related to the infection and without improvement, despite appropriate antibiotics or other treatment) Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no | <del> </del> | |
| 13 | information on the excretion of agents into breast milk. All females of childbearing potential must have a blood | | |
| | test or urine study within 2 weeks prior to registration to rule out pregnancy. | | |
| 14 | | | |
| | Patient Given Copy of Consent: Yes, Date No Having obtained consent and reviewed each of the inclusion/exclusion criteria, I verify this patient is: Eligible Ineligible Date Registered | that | |
| | Signature of Person Completing This Form | | |

Bridging Study Version 5.0 Confidential Page 46 of 52



### APPENDIX 2 Performance Status Criteria

## For patients 16 years of age and older:

| | Karnofsky Performance Scale |
|---|---|
| Percent | cent Description |
| 100 | Normal, no complaints, no evidence of disease. |
| 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 80 | Normal activity with effort; some signs or symptoms of disease. |
| 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| 50 | Requires considerable assistance and frequent medical care. |
| 40 | Disabled, requires special care and assistance. |
| 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 20 | Very sick, hospitalization indicated. Death not imminent. |
| 10 | Moribund, fatal processes progressing rapidly. |
| 0 | Dead |

### For patients less than 16 years of age:

| | Lansky Performance Scale |
|---|---|
| Lansky | Lansky Play Score |
| Score | |
| 100 | Fully active, normal |
| 90 | Minor restrictions in physically strenuous activity |
| 80 | Active, but tires more quickly |
| 70 | Both greater restriction of and less time spent in play activity |
| 60 | Up and around, but minimal active play; keeps busy with quieter activities |
| 50 | Gets dressed but lies around much of the day, no active play but able to |
| | participate in all quiet play and activities |
| 40 | Mostly in bed; participates in quiet activities |
| 30 | In bed; needs assistance even for quiet play |
| 20 | Often sleeping; play entirely limited to very passive activities |
| 10 | No play; does not get out of bed |
| 0 | Unresponsive |



## APPENDIX 3 Response Criteria

#### **Modified RECIST**

### **Complete Remission (CR)**

CR requires that all of the following be present:

- Peripheral Blood Counts
  - $\circ$  ANC count  $> 1.000/\text{mm}^3$
  - o Platelet count > 100.000/mm<sup>3</sup>
  - o Reduced hemoglobin concentration or hematocrit has no bearing on remission status
  - o Leukemic blasts must not be present in the peripheral blood
- Marrow Aspirate and Biopsy
  - Bone marrow biopsy must demonstrate tri-lineage hematopoiesis with maturation of all cell lines.
  - o < 5% blasts
- Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present.

### Morphological Remission (MR)

MR requires that the following be present:

• Patient meets all peripheral blood and bone marrow criteria for CR, except that platelet count is < 100,000/mm<sup>3</sup> but > 50,000/mm<sup>3</sup>

### Minimal Residual Disease (MRD) Negativity

- MRD negativity for ALL requires the following be present:
  - < 0.01% leukemic blasts by flow cytometry
  - o Absence of cytogenetic and/or molecular evidence of disease if applicable
- MRD negativity for AML requires the following be present:
  - < 0.5% leukemic blasts by flow cytometry
  - o Absence of cytogenetic and/or molecular evidence of disease if applicable

### Relapse

Relapse following CR is defined as:

- Peripheral Blood Counts
  - Presence of peripheral blasts. A bone marrow examination must be performed to confirm relapse. However, please note that the date of relapse is the first date at which the relapsed patient had: leukemic blasts in the peripheral blood smear, or >5% blasts in the bone marrow.
- Bone Marrow Aspirate or Biopsy
  - o Presence of more than 5% blasts, not attributable to another cause (i.e. bone marrow regeneration).



# APPENDIX 4 Known and Expected Toxicities of Study Treatment



| | Known I | Risks and Side Effect | s Re | elated to the <u>Clofarabine</u> Incl | ude Tł | nose Which Are: |
|---|---|---|---|---|---|---|
| | ] | Likely | Less Likely | | Rare But Serious | |
| | other places | s in the body | | that can make you feel short | pa | ancreas and which may |
| • | Bloody nos | e | | of breath | ca | ause pain in the |
| • | Fewer white | e blood cells, red | • | Severe rash with redness | ał | odomen (belly) which |
| | blood cells | and platelets in the | | and pain on the palms of the | | an be severe and may |
| | blood | | | hand and soles of the feet | in | crease the blood sugar |
| | o a low m | umber of white | • | Red spots on the skin from | | |
| | blood co | ells can make it | | low platelets | | |
| | | get infections | • | High levels of uric acid in | | |
| | o a low m | umber of red blood | | the blood which could | | |
| | cells car | n make you feel tired | | damage the kidneys | | |
| | and wea | | • | Increased levels of a | | |
| | | umber of platelets | | chemical (creatinine) in the | | |
| | - | you to bruise and | | blood which could mean | | |
| | bleed m | ore easily | | kidney damage | | |

| | Known Risks and Side Effects Related to Cyclophosphamide Include Those Which Are: | | |
|---|---|---|---|
| | Likely | Less Likely | Rare But Serious |
| • | Loss of appetite | Abnormal hormone function which | Heart muscle damage |
| • | Nausea | may lower the level of salt in the blood | which may occur with |
| • | Vomiting | Abdominal pain | very high doses and |
| • | Fewer white blood | • Diarrhea | which may be fatal |
| | cells in the blood. | • Fewer red blood cells and platelets in | Abnormal heart rhythms |
| | o a low number of | the blood | • Damage and scarring of |
| | white blood | <ul> <li>a low number of red blood cells</li> </ul> | lung tissue which may |
| | cells may make | may make you feel tired and weak. | make you short of breath |
| | it easier to get | a to whatteet of placetes may | A new cancer or leukemia |
| | infections. | cause you to bruise and bleed more | resulting from this |
| • | Hair loss | easily. | treatment. |
| • | Decreased ability of | Breeding and installmation of the | Damage or scarring of |
| | the body to fight | urinary bladder | urinary bladder tissue |
| | infection | reserves of decrease monthly periods | Severe allergic reaction |
| • | Absence or | which may be temporary or permanent | which can be life |
| | decrease in the | and which may decrease the ability to | threatening with shortness |
| | number of sperm | have children | of breath, low blood |
| | which may be | • Temporary blurred vision | pressure, rapid heart rate chills and fever |
| | temporary or | Nasal stuffiness with IV infusions | |
| | permanent which may decrease the | JKIII Tusii | • Infertility which is the inability to have children |
| | ability to have | • Darkening of areas of the skin and | madnity to have children |
| | children | finger nails | |
| | Cilitatell | Slow healing of wounds | |
| | | • Infections | |

| Known Risks and Side Effects Related to Etoposide Include Those Which Are: | | |
|---|---|---|
| Likely | Less Likely | Rare But Serious |
| Nausea and vomiting | • Loss of appetite | Damage to the liver |



There also may be other side effects that we cannot predict. Many side effects go away shortly after the drugs are stopped, but in some cases side effects can be serious, long-lasting, or permanent. Other drugs may be given to make side effects less serious and uncomfortable.



### **APPENDIX 5**

### **Bridging Therapy Roadmap**

| Drug | Route | Dosage | Days |
|---|---|---|---|
| Clofarabine | IV over 2 hours | 20 mg/m <sup>2</sup> | 1-5 |
| Etoposide (ETOP) | IV over 2 hours | 100 mg/m <sup>2</sup> | 1-5 |
| Cyclophosphamide (CYCLO) | IV over 30 to 60 mins | $300 \text{ mg/m}^2$ | 1-5 |

### **Drugs Given In This Order:**

Clofarabine 20 mg/m<sup>2</sup> IV over 2 hours followed by

Etoposide 100 mg/m<sup>2</sup> IV over 2 hours followed by

Cyclophosphamide  $300 \text{ mg/m}^2 \text{ IV}$  as a 30-60 minute infusion

| Ht | Wt. | BSA |
|----|--------|------|
| | , , •• | 2011 |

| Date<br>Due | Date<br>Given | Day | Clofarabine | ЕТОР | CYCLO |
|-------------|---------------|------|-----------------|------|-------|
| Due | Given | | mg | mg | mg |
| | | 1 | mg | mg | mg |
| | | 2 | mg | mg | mg |
| | | 3 | mg | mg | mg |
| | | 4 | mg | mg | mg |
| | | 5 | mg | mg | mg |
| | | 6-28 | No Chemotherapy | | |